| PROTOCOL | |
|---|---|
| TITLE: | Letermovir for cytomegalovirus prophylaxis in patients with |
| | hematological malignancies treated with alemtuzumab |
| STUDY NUMBER: | OSU-19289 |
| IND NUMBER: | 147864 |
| TEST PRODUCTS: | NA |
| COMMERICAL PRODUCTS: | Letermovir |
| INDICATION: | Hematologic malignancies treated with alemtuzumab |
| INVESTIGATOR: | John C. Reneau, MD, PhD |
| | 320 West 10 <sup>th</sup> Avenue |
| | A350A Starling Loving Hall |
| | Telephone: 614-688-7942 |
| | Fax: 614-293-7526 |
| | E-mail: john.reneau@osumc.edu |
| Statistician | Ying Huang, MSc |
| | 320 West 10th Avenue |
| | Telephone: 614-688-7591 |
| | Fax: 614-293-7526 |
| | Email: <a href="mailto:ying.huang@osumc.edu">ying.huang@osumc.edu</a> |
| SUPPORT PROVIDED BY: | The Ohio State University |
| | Merck |

1

2

4 5 6

3

7

#### **CONFIDENTIAL**

This is an Ohio State University document that contains confidential information. It is intended solely for the recipient clinical investigator(s) and must not be disclosed to any other party. This material may be used only for evaluating or conducting clinical investigations; any other proposed use requires written consent from Ohio State University.

#### 9 **TABLE OF CONTENTS** 10 Background and Rationale......7 11 1 12 1.1 13 1.1.1 14 1.1.2 1.1.3 15 16 1.2 Alemtuzumab......8 17 1.3 18 1.4 19 2 Objectives......11 20 2.1 21 2.1.1 Primary Objective ......11 22 2.1.2 23 2.1.3 Exploratory Objectives ......11 24 2.2 25 2.2.1 Primary Endpoint ......11 2.2.2 26 27 2.2.3 28 3 29 3.1 Inclusion Criteria ......11 30 3.2 31 3.3 Treatment Plan .......15 32 4.1 33 4.2 Agent Administration......15 34 4.3 35 36 4.4 Concomitant Medications and Supportive Care ......16 37 5 5.1 38 Dose Delays and Modifications......17 5.2 39 40 Calendar of Events ......18 41 6.1

| 42 | 6.2 | Biospecimen Studies and Procedures | |
|---|---|---|---|
| 43 | 6.3 | Source and Timing of Biospecimen Collections | 19 |
| 44 | 6.4 | Storage of Biospecimens | 19 |
| 45 | 7 Crit | teria for Disease Evaluation | 19 |
| 46 | 8 Let | ermovir Information | 19 |
| 47 | 8.1 | Letermovir Description and Mechanism of Action | 19 |
| 48 | 8.2 | Clinical Pharmacology | 20 |
| 49 | 8.3 | Pharmacokinetics and Drug Metabolism | 20 |
| 50 | 8.4 | Preparation, Storage, and Administration: Oral Formulation | 33 |
| 51 | 8.5 | Preparation, Storage, and Administration: Intravenous formulation | 34 |
| 52 | 8.6 | Non Clinical Toxicology | 36 |
| 53 | 8.6 | .1 Carcinogenesis, Mutagenesis, Impairment of Fertility | 36 |
| 54 | 8.6 | .2 Animal Toxicology and Pharmacology | 36 |
| 55 | 8.7 | Clinical Studies | 36 |
| 56 | 8.8 | Adverse Events | 41 |
| 57 | 9 Re | gulatory and Reporting Requirements | 43 |
| 58 | 9.1 | Adverse Events (AEs) | 43 |
| 59 | 9.2 | Serious Adverse Events (SAEs) | 44 |
| 60 | 9.3 | Noncompliance | 44 |
| 61 | 9.4 | Serious Noncompliance | 45 |
| 62 | 9.5 | Reporting to the OSU IRB | 45 |
| 63 | 9.6 | Reporting to the sponsor4 | |
| 64 | 9.7 | 9.7 Reporting to the FDA | |
| 65 | 9.8 | Timeframe for Reporting Required Events | 46 |
| 66 | 9.9 | Overdose | 47 |
| 67 | 9.10 | Pregnancies | 47 |
| 68 | 9.11 | Data and safety monitoring | 47 |
| 69 | 9.1 | 1.1 Data Submission | 48 |
| 70 | 9.1 | 1.2 Auditing | 48 |
| 71 | 9.12 | Ethical Considerations | 48 |
| 72 | 9.13 | Retention of records | 48 |
| 73 | 10 5 | Statistical Methods | 48 |
| 74 | 10.1 | Study Design and Sample Size Justification | 48 |
| 75 | 10.2 | Analysis of Primary Objective | 49 |
| 76 | 10.3 | Analysis of Secondary Objectives | 49 |

| | | | pp10104. 201 002020 |
|---|---|---|---|
| 77 | 10.4 | Analysis of Exploratory Objectives | 50 |
| 78 | 11 F | References | 50 |
| 79 | 12 | Appendices | 54 |
| 80<br>81 | 12.1<br>Forui | CMV Disease Definitions Working Group of the Cytomegalovirus Drum54 | ug Development |
| 82 | 12.2 | Eastern Cooperative Oncology Group Performance Status Scale | 56 |
| 83 | 12.3 | Child-Pugh Classification of liver disease | 57 |
| 84 | | | |
| 85 | | | |

# **TRIAL SUMMARY**

| TITLE | Letermovir for cytomegalovirus prophylaxis in patients with |
|---|---|
| | hematological malignancies treated with alemtuzumab |
| PHASE | |
| OBJECTIVES | Primary Objective |
| | 1. To estimate the rate of CMV reactivation in patients treated with letermovir at 3 months after completion of alemtuzumab therapy. |
| | letermovir at 3 months after completion of alemitizumab therapy. |
| | Secondary Objectives |
| | To evaluate the tolerability of letermovir in combination with |
| | alemtuzumab. |
| | 2. To evaluate the efficacy of letermovir for the prevention of clinically |
| | significant CMV disease. |
| | 4. To estimate the overall survival of patients in the study population |
| STUDY DESIGN | Single center, single arm, non-randomized |
| KEY ELIGIBILITY | Inclusion Criteria |
| CRITERIA | 1. Confirmed diagnosis of any lymphoid malignancy including, but not limited to, T- or B-PLL, CLL, PTCL, CTCL, Sézary syndrome, or |
| | LGLL. |
| | 2. Intent to treat with alemtuzumab (monotherapy or in combination |
| | with chemotherapy). |
| | Confirmed seropositivity for CMV IgG |
| | 4. Confirmed lack of active CMV infection as evidenced by CMV DNA |
| | PCR ≤ 200 IU/mL and no clinical evidence of CMV disease within 14 |
| | days of first letermovir dose. |
| | 5. Age ≥18 years old |
| | 6. Able to provide informed consent |
| | 7. Life expectancy >4 months 8. ECOG performance status ≤3 |
| | 9. Highly unlikely to become pregnant or impregnate a partner (post- |
| | menopausal, sterile, abstinence, or adequate contraceptive method) |
| | Exclusion Criteria |
| | 1. History of confirmed CMV disease within 1 year of study entry. |
| | 2. History of prior allogeneic hematopoietic stem cell transplant within 6 months of enrollment. Allogeneic transplant more than 6 months |
| | prior to enrollment is allowed as long as the subject is off |
| | immunosuppression without active GVHD. |
| | 3. End stage renal disease with creatinine clearance < 10 mL/min |
| | 4. Severe hepatic impairment defined as Child-Pugh class C OR AST |
| | or ALT > 5 x ULN OR serum total bilirubin > 2.5 x ULN. |
| | 5. Both moderate hepatic insufficiency AND moderate renal |
| | insufficiency defined as Child Pugh Class B AND creatinine clearance |
| | less than 50 mL/min |
| | <ul><li>6. Cytopenias are NOT an exclusion criteria</li><li>7. Received antiviral medications with activity against CMV or</li></ul> |
| | contraindicated medication within specified windows (see Section 3.2 |
| | for details) |
| | 8. Received cidofovir, CMV hyper-immune globulin, or an |
| | investigational anti CMV agent within 30 days. |

| | 11 to 7 pp 10 to 4. 201 052020 |
|---|---|
| STATISTICS | 9. Infection or underlying disease necessitating ongoing use of prohibited medications (Section 4.4). 10. Suspected or known hypersensitivity to active or inactive ingredients of letermovir formulations 11. Active HIV, hepatitis B, or hepatitis C infection (see section 3.2 for exceptions) 12. Pregnant, breastfeeding, or expecting to conceive. 13. Expecting to donate eggs or sperm 14. Current or recent participation in a study with an unapproved investigational compound. 15. Previous participation in a study using letermovir. 16. Any condition which might interfere with subjects participation as judged by investigator. The primary objective of this single center, single arm phase II study is to determine the efficacy of letermovir prophylaxis in PLL, CLL, PTCL or CTCL patients treated with alemtuzumab. The efficacy will be measured through the CMV reactivation rate during letermovir prophylaxis (3 months after completion of alemtuzumab therapy). All eligible patients who receive any letermovir will be included in the tolerability analysis, and all patients who receive ≥90% of planned letermovir doses are evaluable for the efficacy analysis. Fleming's two-stage design will be used with the following parameters: • Null hypothesis: CMV reactivation rate of 30% or higher is not acceptable (70% safety rate) • Alternative hypothesis: CMV reactivation rate of 10% or less is acceptable (90% safety rate) With a one-sided type I error rate of 5% and 85% power, Fleming's two-stage design allows a first-stage analysis after the first 14 patients are enrolled and evaluated: • If ≥4 CMV reactivations, trial will terminate due to futility • If 0 CMV reactivations, trial will terminate due to efficacy • If at least 24 of 28 enrolled patients are CMV free, we will conclude the regimen effective |
| | To account for the possibility that some patients will not be evaluable, |
| | we will allow a 5% over-accrual for a total target enrollment of 30. |
| TOTAL NUMBER OF SUBJECTS | 14 to 30 depending upon results of interim analysis. |
| ESTIMATED ENROLLMENT | Stage 1: 10 months from first patient enrolled Stage 2: 20 months from first patient enrolled |
| PERIOD | · |
| ESTIMATED STUDY DURATION | Stage 1: 17 months from first patient enrolled Stage 2: 27 months from first patient enrolled |

#### 1 BACKGROUND AND RATIONALE

# 89 1.1 Mature T-cell Lymphomas

- 90 Approximately 10-15% of non-Hodgkin lymphomas (NHL) are derived from mature (i.e. post-
- 91 thymic) T lymphocytes [1]. The heterogeneity of these lymphomas and poor understanding of
- 92 their pathogenesis continue to impede their classification and the development of novel
- 93 therapeutic strategies.

88

94

120

## 1.1.1 Peripheral T-cell Lymphoma

- 95 The most common subtype of peripheral T-cell lymphoma (PTCL) lacks any distinguishing
- 96 characteristics and is designated by the World Health Organization as "PTCL, not otherwise
- 97 specified (PTCL, NOS)" [1, 2]. While the development of combination immunochemotherapy
- 98 (e.g. "R-CHOP") has led to significant survival benefits in B-cell NHL, the PTCLs are associated
- 99 with inferior responses to therapy and overall survival [3]. In fact, the vast majority of PTCL
- patients will ultimately succumb to their disease, most within a few years of diagnosis [1, 2, 4].
- Novel therapeutic strategies are needed if improved outcomes are to be achieved. The
- 102 observation that PTCL incidence rates are increasing faster than almost any other subgroup of
- 103 NHL further heightens this sense of urgency [5, 6].

# 104 1.1.2 Cutaneous T-cell Lymphoma

- 105 Primary cutaneous T-cell lymphoma (CTCL), of which the two most common forms are mycosis
- 106 fungoides (MF) and Sézary syndrome (SS), predominantly involves the skin. Most CTCL
- patients present with limited-stage disease that is confined to the skin (i.e. patches or plaques)
- and are managed with topical therapies. In contrast, patients with advanced-stage disease with
- significant blood, nodal or visceral organ involvement are managed with systemic therapies [7].
- 110 A variety of single agent or combination chemotherapy regimens are utilized, as there is no
- 111 standard of care for these patients. Therefore, the National Comprehensive Cancer Network
- 112 (NCCN) guidelines endorse these agents or participation in a clinical trial as first-line therapy in
- these patients. Median overall survival for patients with stage IV disease ranges from 1.4-3.8
- 114 years, depending upon the extent of blood, nodal or visceral organ involvement [8]. Five FDA
- approved agents are currently available for CTCL patients failing at least one prior therapy.
- including bexarotene, vorinostat, romidepsin, brentuximab vedotin (for CD30 positive disease),
- and mogamulizumab. These agents are associated with overall response rates of 28-56% [9-15]
- with generally short duration of response. Despite the use of these novel agents, the long term
- outlook for most CTCL patients remains grim.

# 1.1.3 T-cell Prolymphocytic Leukemia

- 121 T-cell prolymphocytic leukemia (T-PLL) is a rare T-cell malignancy most often presenting in
- adult males[16]. While most presentations of this disease are acute, a minority of patients will
- not require treatment immediately. There is a limited response to conventional chemotherapy
- 124 with alkylating agents or anthracyclines, with a median overall survival (OS) of 7 months in
- historical series [16, 17]. In the absence of a clinical trials, patients should be offered
- 126 alemtuzumab as front line therapy. Alemtuzumab has a high overall response rate >80% in the
- front line setting [18] and 51-76% in the relapsed setting [19-22]. Even with high response rates,
- relapse is common in the absence of consolidative therapy. Allogeneic hematopoietic stem cell

- transplantation is frequently recommended as consolidation therapy with resulted prolongation
- of overall survival and cure in a minority of cases [23-26]

#### 1.2 Alemtuzumab

131

- 132 Alemtuzumab is a humanized IgG1 kappa monoclonal antibody directed against the CD52
- antigen, which is mostly expressed by B- and T-lymphocytes. Clinical activity of alemtuzumab
- has been evaluated in multiple lymphoid malignancies including peripheral T cell lymphoma
- 135 (PTCL), mycosis fungoides (MF), Sézary syndrome (SS), T-cell prolymphocytic leukemia (T-
- 136 PLL), and chronic lymphocytic leukemia (CLL)[27].
- 137 In the relapsed setting, alemtuzumab monotherapy results in 36% overall response rate (ORR)
- with 21% complete response rate (CRR) in PTCL [28]. Patients with MF/SS have an ORR
- ranging from 55% to 100% with an average ORR of 65% [29]. Patients with erythrodermic MF or
- 140 SS have significantly better responses (ORR 85-100%) even with lower doses of alemtuzumab
- therapy[30, 31]. Alemtuzumab is considered standard front line therapy for symptomatic T-PLL
- 142 (NCCN guidelines) with ORR of 51-76% and CRR of 40-60% [21, 22]. Alemtuzumab has also
- been used in combination with various chemotherapeutic agents in the front line and relapsed
- setting in these diseases including CHOP (cyclophosphamide, doxorubicin, vincristine, and
- prednisone), EPOCH (etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin),
- and pentostatin [32-34]. Efficacy is improved with these combinations, but also results in
- 147 cumulative toxicities.
- In general, therapy with alemtuzumab is well tolerated, but cytomegalovirus (CMV) reactivation
- and other infectious complications remain a significant barrier to more widespread clinical use.
- 150 In clinical trials where data is available, reported rates of CMV reactivation average 30% (see
- 151 Table 1).

152

# 1.3 Cytomegalovirus

- 153 Infection with human cytomegalovirus (CMV) is relatively frequent in the human population with
- a seroprevalence ranging from 45-100% [35]. Following initial exposure, the virus establishes a
- lifelong latent infection that can periodically reactivate with shedding of infectious virus, although
- this rarely results in a clinically significant infection in healthy individuals. In contrast,
- 157 reactivation is responsible for significant mortality and morbidity in immunocompromised
- patients [35]. CMV replication involves the cleaving of concatameric genomic viral DNA and the
- packaging of each genome into preformed viral capsids. This process is mediated by the CMV-
- terminase complex (UL51, UL56, and UL89) [36].
- 161 Risk factors associated with CMV reactivation include seropositivity of the recipient while
- undergoing therapy immunosuppressive therapy with autologous or allogeneic transplant or
- drugs like high dose steroids or alemtuzumab. Clinical manifestations include interstitial
- pneumonitis, encephalitis, retinitis, fevers, hepatitis, hemorrhagic cystitis and diarrhea [37].
- 165 Current management focuses on reduction in immunosuppression and initiation of antiviral
- therapies including ganciclovir, cidofovir, foscarnet, and valganciclovir [37, 38]. Use of these
- agents, while necessary, carries significant side effect profiles including marrow suppression
- and nephrotoxicity. Furthermore, the development of antiviral resistance via mutations to CMV
- 169 UL97 or UL54 genes limits the available agents effective against CMV [38]. Antiviral drug
- 170 resistance should be suspected in patients who fail to improve (i.e., >1 log<sub>10</sub> increase in CMV

- 171 DNA levels in blood or serum) after 2 weeks of appropriately dosed antiviral therapy [38].
- 172 Although the incidence of drug resistant CMV remains low (0-8%)[39, 40], it can still pose
- significant challenges to treatment when it occurs. Therefore, novel therapies to reduce the risk
- of CMV reactivation are needed in order to avoid serious side effects of antiviral therapies and
- to avoid drug resistance to these agents.
- 176 A review of published studies using alemtuzumab in the target patient population for this trial is
- 177 summarized in Table 1. This shows that the CMV reactivation rate in this patient population is
- 178 ~30%.

179

180

# Table 1: Reported rates of CMV reactivation with alemtuzumab in target patient population

| Ref | Population | CMV<br>Reactivation<br>(n) | Total<br>Patients<br>(n) | Reactivation<br>Rate | CMV<br>Prophy* | Chemo<br>Combination | Front<br>Line<br>Therapy | Relapsed<br>Therapy |
|---|---|---|---|---|---|---|---|---|
| [34] | PTCL, T-<br>PLL, T-LGL,<br>T-ALL, MF | 9 | 24 | 38% | Y | Υ | Υ | Y |
| [41] | HTLV+<br>ATLL | 29 | 29 | 100% | Υ | N | Υ | Υ |
| [42] | PTCL | 5 | 20 | 25% | N | Υ | Υ | N |
| [43] | PTCL | 5 | 41 | 12% | N | Υ | Υ | N |
| [32] | PTCL | 7 | 20 | 35% | N | Υ | Υ | N |
| [44] | PTCL | 12 | 38 | 32% | N | Υ | Υ | Υ |
| [33] | PTCL | 16 | 31 | 52% | N | Υ | Υ | N |
| [45] | T-PLL | 13 | 21 | 62% | N | Υ | Υ | N |
| [46] | PTCL, T-<br>ALL | 6 | 13 | 46% | N | Υ | Υ | Υ |
| [47] | PTCL | 8 | 15 | 53% | N | Υ | Υ | N |
| [48] | PTCL | 8 | 24 | 33% | N | Υ | N | Υ |
| [49] | SS | 3 | 5 | 60% | N | Υ | N | Υ |
| [30] | SS | 3 | 14 | 21% | N | N | Υ | Υ |
| [50] | CTCL | 10 | 39 | 26% | N | N | Υ | Υ |
| [51] | T-LGL | 6 | 13 | 46% | N | N | Υ | Υ |
| [20] | CLL, PLL,<br>CTCL,<br>PTCL, T-<br>LGL, MCL,<br>HCL | 15 | 78 | 19% | N | N | Y | Y |
| [52] | SS | 2 | 5 | 40% | N | N | Υ | Υ |
| [21] | T-PLL | 3 | 76 | 4% | N | N | Υ | Υ |
| [28] | PTCL | 6 | 14 | 43% | N | N | N | Υ |
| [53] | CLL, PLL | 5 | 34 | 15% | N | N | N | Υ |
| [54] | MF, SS | 0 | 10 | 0% | N | N | N | Υ |
| [55] | PTCL, CTCL | 1 | 10 | 10% | N | N | N | Υ |
| [56] | MF, SS | 1 | 8 | 13% | N | N | N | Υ |
| [57] | MF, SS | 4 | 22 | 18% | N | N | N | Υ |
| [58] | MF, SS | 0 | 18 | 0% | N | N | N | Υ |

| Ref | Population | CMV<br>Reactivation<br>(n) | Total<br>Patients<br>(n) | Reactivation<br>Rate | CMV<br>Prophy* | Chemo<br>Combination | Front<br>Line<br>Therapy | Relapsed<br>Therapy |
|---|---|---|---|---|---|---|---|---|
| [59] | SS | 3 | 6 | 50% | N | N | N | Υ |
| [60] | PTCL | 10 | 20 | 50% | NR | Υ | Υ | N |
| [61] | PTCL | 5 | 16 | 31% | NR | Υ | N | Υ |
| [62] | PTCL | 1 | 10 | 10% | NR | Υ | N | Υ |
| [18] | T-PLL | 2 | 9 | 22% | NR | N | Υ | N |
| [22] | T-PLL | 1 | 39 | 3% | NR | N | Υ | Υ |
| [19] | T-PLL | 1 | 15 | 7% | NR | N | N | Υ |
| [63] | SS | 6 | 13 | 46% | NR | N | N | Υ |
| [64] | SS | 1 | 1 | 100% | NR | N | N | Υ |
| [65] | SS | 3 | 6 | 50% | NR | N | NR | NR |
| [66] | NHL, PTCL,<br>AML, ALL,<br>MDS, AA | 66 | 180 | 37% | Variable | Y | Y | Y |

TOTAL 276 937 29%

\*CMV prophylaxis defined as planned routine use of: ganciclovir (any dose), valganciclovir (any dose), foscarnet (any dose), acyclovir (>3200 mg by mouth per day or >25 mg/kg IV per day), valacyclovir (>3000 mg by mouth per day), or famciclovir (>1500 mg by mouth daily).

Abbreviations: AA = aplastic anemia, ALL = T-cell acute lymphoblastic leukemia, AML = acute myeloid leukemia, ATLL = adult T-cell leukemia/lymphoma, CLL = chronic lymphocytic leukemia, CMV = cytomegalovirus, CTCL = cutaneous T-cell lymphoma, HCL = hairy cell leukemia, HTLV = human T-lymphotropic virus, MCL = mantle cell lymphoma, MDS = myelodysplastic syndrome, MF = mycosis fungoides, N = no, NHL = non-Hodgkin lymphoma, NR = not reported, PLL = prolymphocytic leukemia, Prophy = prophylaxis, PTCL = peripheral T cell lymphoma, SS = Sézary syndrome, T-LGL = T-cell large granular lymphocytic leukemia, Y = yes

#### 1.4 Letermovir

181

182

183

184

- Letermovir is a highly potent anti-CMV agent recently FDA approved for anti-CMV prophylaxis post-transplant based on the results of a recent randomized phase 3 trial [67]. Letermovir inhibits CMV replication by binding components of the terminase complex resulting in impaired cleavage and packaging of viral DNA into capsids [68, 69].
- In the trial leading to FDA approval, 565 CMV seropositive patients without detectable CMV
- 187 DNA at baseline undergoing allogeneic hematopoietic stem cell transplantation were
- randomized to receive letermovir prophylaxis or placebo through week 14 after transplantation.
- 189 Patients treated with letermovir experienced a statistically significant decrease in clinically
- significant CMV infection compared to placebo (37.5% vs 60.6%, P<0.001). Additionally, the
- 191 frequency and severity of adverse events were statistically similar between the two groups
- 192 overall. Patients in the letermovir group may have experienced slightly higher rates of nausea
- and vomiting, peripheral edema, and atrial fibrillation. Importantly, the use of letermovir
- 194 prophylaxis was associated with a trend toward lower all-cause mortality compared to placebo
- in this trial and this was confirmed in a post hoc analysis of survival [70].

- 196 Based on these data and the high rate of CMV reactivation following alemtuzumab therapy, we
- 197 propose the following phase 2 clinical trial of letermovir prophylaxis in patients with hematologic
- 198 malignancies receiving alemtuzumab.

#### 2 OBJECTIVES AND ENDPOINTS

# 200 2.1 Objectives

199

202

203

205

210

213

#### 201 **2.1.1 Primary Objective**

1. To estimate the rate of CMV reactivation in patients treated with letermovir at 3 months after completion of alemtuzumab therapy.

## 204 **2.1.2 Secondary Objectives**

- 1. To evaluate the tolerability of letermovir in combination with alemtuzumab
- To evaluate the efficacy of letermovir for the prevention of clinically significant CMV
   disease
- 208 3. To estimate the overall survival of patients in the study population

# 209 **2.1.3 Exploratory Objectives**

1. To evaluate mechanisms of antiviral resistance in letermovir prophylaxis failures.

## 211 **2.2 Endpoints**

## 212 **2.2.1 Primary Endpoint**

1. CMV reactivation as defined in section 10.2.

#### 214 2.2.2 Secondary Endpoints

- Adverse events (AEs) using NCI Common Terminology Criteria for Adverse Events
   (CTCAE) version 5.
- Development of CMV disease per the Disease Definitions Working Group of the
   Cytomegalovirus Drug Development Forum [71] (Appendix 12.1)
- 3. Overall survival as defined in section 10.3

#### 220 **2.2.3 Exploratory Endpoints**

Genotyping to evaluate mutations in CMV terminase complex genes (UL51, UL56, UL89) [72-79]

#### 223 3 PATIENTS AND METHODS

#### 224 3.1 Inclusion Criteria

- Confirmed diagnosis of any lymphoid malignancy including, but not limited to, T-cell or
   B-cell prolymphocytic leukemia, chronic lymphocytic leukemia, peripheral T-cell
- lymphoma, cutaneous T-cell lymphoma, Sézary syndrome, or large granular lymphocytic leukemia.

- 229 Intent to treat with alemtuzumab. Monotherapy or combination with chemotherapy is 230 allowed. 231 3. Confirmed seropositivity for CMV IgG (≥0.7 U/mL) within 1 year of first letermovir dose. 232 Confirmed lack of active CMV infection as evidenced by CMV DNA PCR ≤ 200 IU/mL and no clinical evidence of CMV disease within 14 days of first letermovir dose. 233 234 5. Age ≥18 years old 235 6. Able to provide informed consent. 236 7. Life expectancy >4 months 237 8. Eastern Cooperative Oncology Group (ECOG) performance status ≤3 (Appendix 12.2) 238 9. Highly unlikely to become pregnant or impregnate a partner by meeting at least one of 239 the following: 240 a. A female subject who is not of reproductive potential is eligible without requiring 241 the use of contraception. A female subject who is not of reproductive potential is 242 defined as one who: 243 i. has reached natural menopause (defined as 6 months of spontaneous 244 amenorrhea with serum follicle-stimulating hormone [FSH] levels in the 245 postmenopausal range as determined by the local laboratory, or 12 246 months of spontaneous amenorrhea) 247 OR 248 ii. is 6 weeks post-surgical bilateral oophorectomy with or without 249 hysterectomy 250 OR 251 iii. has undergone bilateral tubal ligation. Spontaneous amenorrhea does not include cases for which there is an underlying disease that causes 252 253 amenorrhea (e.g., anorexia nervosa). 254 b. A male subject who is not of reproductive potential is eligible without requiring the 255 use of contraception. A male subject who is not of reproductive potential is 256 defined as one whom has undergone a successful defined as: 257
  - - i. microscopic documentation of azoospermia

258 259

260 261

262

263 264

265

266

267

268 269

- ii. a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy
- c. A male or female subject who is of reproductive potential agrees to true abstinence or to use (or have their partner use) an acceptable method of birth control starting from the time of consent through 90 days after the last dose of study therapy. True abstinence is defined as abstinence in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., abstinence only on certain calendar days, abstinence only during ovulation period, use of symptothermal method, use of post-ovulation methods) and withdrawal are not acceptable methods of contraception. Acceptable methods of birth control are:
  - i. intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, and vasectomy OR use of appropriate double barrier

contraception. Hormonal contraceptives (e.g., birth control pills, transdermal patch, or injectables) are also acceptable.

#### 3.2 Exclusion Criteria

273

275

276

277

278

281

284

285 286

287

288

289 290

291

292

293

294

295

296

297

298

299

300

301

302

303

304

- 1. History of confirmed CMV disease within 1 year of study entry.
  - History of prior allogeneic hematopoietic stem cell transplant within 6 months of trial enrollment. Subjects who have undergone allogeneic transplant more than 6 months prior to enrollment are eligible as long as the subject is off immunosuppression without active GVHD.
- 3. End stage renal disease with creatinine clearance < 10 mL/min as defined by Cockcroft-Gault equation using serum creatinine within 7 days of enrollment
  - a. Creatinine clearance (males) =  $\frac{\text{(Weight in kg)(140-age)}}{\text{(72)(creatinine in mg/dL)}}$
- b. Creatinine clearance (females) =  $\frac{\text{(Weight in kg)(140-age)}}{\text{(72)(creatinine in mg/dL)}} * 0.85$
- 4. Severe hepatic impairment defined as:
  - a. Child-Pugh class C (see appendix 12.2) within 7 days of enrollment
  - b. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN.

<u>Note:</u> Subjects who meet this exclusion criterion may, at the discretion of the investigator, have one repeat testing done. If the repeat value does not meet this criterion, they may continue in the screening process. Only the specific out of range value should be repeated (not the entire panel).

- 5. Both moderate hepatic insufficiency AND moderate renal insufficiency:
  - a. Moderate hepatic insufficiency is defined as Child Pugh Class B (see Appendix 12.2)
  - b. Moderate renal insufficiency is defined as a creatinine clearance less than 50 mL/min, as calculated by the Cockcroft-Gault equation (as above)
- Cytopenias are NOT an exclusion criteria in this trial as cytopenias are common in this
  patient population and letermovir has no known adverse effects on blood counts.
  Patients will be treated per institutional standard of care with as needed transfusions and
  growth factor support.
- 7. Received any of the following drugs within 7 days of enrollment or plans to receive any of the following during the study:
  - a. ganciclovir
  - b. valganciclovir
  - c. foscarnet
- d. acyclovir (at doses > 3200 mg PO per day or > 25 mg/kg IV per day)
- e. valacyclovir (at doses > 3000 mg PO per day)
- f. famciclovir (at doses > 1500 mg PO per day)
- 308 g. Cyclosporine A

309 h. Pimozide 310 Ergot alkaloids (ergotamine and dihydroergotamine) 311 j. Atorvastatin at doses greater than 20 mg daily (see Table 5) 312 8. Received any of the following within 30 days prior to enrollment 313 a. cidofovir 314 b. CMV hyper-immune globulin 315 c. Any investigational CMV antiviral agent/biologic therapy 316 9. Infection or underlying disease necessitating ongoing use of prohibited medications 317 (Section 4.3). 318 10. Suspected or known hypersensitivity to active or inactive ingredients of letermovir 319 formulations 320 11. Positive at the time of screening for: 321 a. HIV with CD4 count <350. If HIV positive, must remain on antiretroviral therapy 322 that is not anticipated to interact with letermovir throughout study. 323 b. Hepatitis B surface antigen or core antibody positivity associated with detectable 324 viral load. For any patient with serologic evidence of prior infection but 325 undetectable viral load, viral load and surface antigen will be monitored every 2 326 weeks. Those with evidence of reactivation (detectable viral load) will be treated 327 with entecavir or lamivudine. Upon resolution of detectable viral load, the patient 328 will be allowed to continue on trial assuming adequate liver function as defined 329 above. Alternatively, patients may be put on prophylactic entecavir or lamivudine 330 to prevent hepatitis B reactivation at the investigators discretion. 331 c. Hepatitis C if no prior or current curative antiviral therapy. For those currently on 332 curative antiviral therapy, they will be allowed on trial if HCV quantitation is below 333 the limit of detection and adequate liver function as above. 334 12. Pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time 335 of consent through 90 days after the last dose of study therapy. 336 13. Expecting to donate eggs or sperm starting from the time of consent through 90 days 337 after the last dose of study therapy. 338 14. Currently participating or has participated in a study with an unapproved investigational 339 compound or device within 28 days, or 5X half-life of the investigational compound 340 (excluding monoclonal antibodies), whichever is longer, of initial dosing on this study. 341 Subjects previously treated with a monoclonal antibody will be eligible to participate after 342 a 28-day washout period. 343 15. Previous participation in a study using letermovir. 344 16. Has a history or current evidence of any condition, therapy, lab abnormality, or other 345 circumstance that might confound the results of the study, interfere with the subject's 346 participation for the full duration of the study, or would be put at undue risk as judged by the investigator, such that it is not in the best interest of the subject to participate in this 347 348 study

## 3.3 Screening Procedures

349

356

358

- 350 Patients may be screened for study entry when the determination has been made by the
- 351 treating physician that they need therapy with alemtuzumab. Application to receive
- 352 alemtuzumab for compassionate use would be started by the treating physician team, as per
- standard of care, while patient is being screened for trial. Application for compassionate use of
- alemtuzumab can be accessed here: <a href="https://www.campathproviderportal.com">https://www.campathproviderportal.com</a>.

#### 355 4 TREATMENT PLAN

#### 4.1 Premedication Administration

No premedication is necessary for letermovir.

# 4.2 Agent Administration

- Letermovir will be administered at 480 mg by mouth daily starting up to two weeks after the first
- 360 administration of alemtuzumab. Treatment will continue for 3 months after the last dose of
- 361 alemtuzumab is given.
- 362 If for any reason, the subject is unable to take the oral formulation of letermovir for an extended
- period of time, the intravenous (IV) formulation of letermovir may be use. Simultaneous use of
- 364 IV and oral study therapy is not allowed. The IV formulation should be switched to oral study
- therapy (i.e., at the next planned dose) as soon as such subjects are able to swallow and/or the
- 366 condition necessitating the use of the IV formulation resolve.
- 367 Study therapy with letermovir may begin as early as the first day of alemtuzumab infusion to no
- 368 later than 14 days after the first alemtuzumab infusion, once the subject is determined to be
- 369 negative for active CMV infection as outlined in the inclusion criteria. Letermovir should continue
- 370 through 90 days after the final planned alemtuzumab infusion.
- 371 Study therapy should be administered at the same time each day. Tablets are to be swallowed
- 372 whole (i.e., no crushing or chewing the tablet is allowed). Study therapy may be administered
- 373 with or without food.
- 374 If a subject misses a dose, the missed dose should be given as soon as possible during the
- 375 same day. If more than 18 hours have gone by after the regular dosing time, then the missed
- dose should be skipped and the normal dosing schedule should be resumed. The next dose
- should not be doubled in order to "make up" what has been missed.
- 378 Study therapy can be administered with or without food. Subjects must avoid consumption of
- 379 grapefruit, Seville oranges or their respective juices, and other quinine-containing drinks or food
- during the trial from 2 weeks prior to study drug administration until 72 hours after the final
- 381 administration of study drug.

#### 4.3 Rationale for Dose Selection

- 383 Please refer to the letermovir package insert for further details of preclinical data and study
- 384 results in humans.

- Letermovir belongs to a new class of anti-CMV agents which have a different mechanism of
- action compared to currently available drugs for the treatment of CMV infection. By inhibiting the
- viral terminase complex, the drug plays a key role in cleavage and packaging of genomic virus
- 388 DNA into provirions.
- 389 Letermovir is anticipated to be efficacious based on both the *in vitro* potency of letermovir as
- well as its *in vivo* efficacy for CMV prophylaxis in a Phase III trial in allogeneic hematopoietic
- 391 stem cell transplantation (HSCT) recipients [67]. In this trial, 565 CMV seropositive patients
- 392 without detectable CMV DNA at baseline undergoing allogeneic HSCT were randomized to
- 393 receive letermovir prophylaxis (480 mg daily or 240 mg daily or patients concomitantly receiving
- 394 CsA) or placebo through week 14 after transplantation. Patients treated with letermovir
- 395 experienced a statistically significant decrease in clinically significant CMV infection compared
- to placebo (37.5% vs 60.6%, P<0.001). Additionally, the frequency and severity of adverse
- events were statistically similar between the two groups overall. Patients in the letermovir group
- may have experienced slightly higher rates of nausea and vomiting, peripheral edema, and
- 399 atrial fibrillation.

407

408

415

- 400 Based on all available safety data, letermovir efficacy in the Phase II and III studies, and the
- 401 exposure-response data, this study will use a dose of 480 mg daily. Patients who have had
- 402 allogeneic transplant within 6 months prior to trial enrollment and patients receiving cyclosporine
- 403 A (CsA) are excluded; phase I studies have demonstrated that co-administration of letermovir
- 404 with CsA increases letermovir exposure ~3 fold. Patients who have undergone allogeneic
- 405 transplant more than 6 months prior to enrollment are eligible as long as the subject is off
- immunosuppression without active GVHD.

# 4.4 Concomitant Medications and Supportive Care

#### Allowed Medications/Therapies

- The following medications/therapies are **allowed** in this study:
- Standard antimicrobial prophylaxis (e.g., levofloxacin for bacteria, fluconazole/ 411 voriconazole/posaconazole for fungi)
- Acyclovir, valacyclovir, or famciclovir for prophylaxis of herpes simplex virus (HSV) or
   varicella zoster virus (VZV) infections at doses no greater than prohibited doses of these
   medications (see below)

#### Prohibited Medications/Therapies

- The following medications/therapies are **prohibited** in this study:
- Antiviral drugs or therapies for prevention/treatment of CMV, including but not limited to:
- 418 ganciclovir
- 419 valganciclovir
- 420 foscarnet
- 421 cidofovir
- acyclovir (at doses > 3200 mg PO per day or > 25 mg/kg IV per day)

423 valacyclovir (at doses > 3000 mg PO per day) 424 • famciclovir (at doses > 1500 mg PO per day) 425 • CMV hyper-immune globulin 426 any investigational CMV antiviral agent/biologic therapy 427 CMV vaccine 428 Investigational Agents 429 Investigational agents are not permitted with the following exceptions: (1) Investigational 430 chemotherapy regimens involving approved agents and (2) investigational antimicrobial 431 regimens involving approved antibacterial/antifungal/antiviral agents. 432 Other Agents: 433 Cyclosporine A 434 Pimozide 435 Ergot alkaloids (ergotamine and dihydroergotamine) Atorvastatin at doses greater than 20 mg daily (see Table 5) 436 Medications/Therapies to be Administered with Caution 437 438 Preclinical studies suggest MK-8228 acts as a weak to moderate inhibitor of cytochrome 439 (CYP)3A4, CYP2C8, CYP2B6 and the transporters OATP1B1 and OATP1B3. It is therefore 440 possible that MK-8228 may increase the exposure of co-administered drugs whose primary 441 route of clearance involves these enzymes or transporters. Please see Table 5 (section 8.3) for a list of potentially clinically significant drug interactions. 442 TOXICITIES, DOSE DELAYS, AND DOSE MODIFICATIONS 443 444 The NCI Common Terminology Criteria for Adverse Events (CTCAE) v5 will be used to grade 445 adverse events. 446 Subjects enrolled in this study will be evaluated clinically and with standard laboratory tests 447 before and at regular intervals during their participation in this study as specified in Study Calendar & Evaluations. 448 449 Subjects will be evaluated for adverse events (all grades), serious adverse events, and adverse 450 events requiring study drug interruption or discontinuation as specified in Study Calendar & 451 Evaluations (section 6). 452 5.1 Dose Delays and Modifications 453 Dose modifications are not allowed on trial. 454 5.2 Protocol Therapy Discontinuation

Subjects may withdraw consent at any time for any reason or be dropped from the trial at the

discretion of the investigator should any untoward effect occur. In addition, a subject may be

455

withdrawn by the investigator or the Sponsor if enrollment into the trial is inappropriate, the trial plan is violated, or for administrative and/or other safety reasons.

459 A subject <u>must</u> be discontinued from the trial for any of the following reasons:

- CMV reactivation as defined in section 10.2 at any time during the study period, study therapy will be discontinued and the subject may be treated according to the local standard of care (outside the context of the study). In this setting, any of the prohibited anti-CMV medications (outlined in section 4.4) may be used.
- The subject becomes pregnant during the study
- The subject's investigator feels it is in the best interest of the subject to discontinue.
- A subject may be discontinued from therapy for any of the following reasons:
  - Any AE/SAE assessed by the physician investigator as possibly or probably related to study therapy. Investigator may continue the subject in the trial if it is deemed to be in the best interest of the subject to stay on study therapy.
  - Failure to comply with the dosing, evaluations, or other requirements of the trial.
  - The subject has a medical condition or personal circumstance which, in the opinion of the investigator and/or Sponsor, places the subject at unnecessary risk through continued participation in the trial or does not allow the subject to adhere to the requirements of the protocol.

#### 6 STUDY EVALUATIONS

#### 6.1 Calendar of Events

460

461 462

463

464

465

467

468

469

470

471

472

473 474

475

| Cycle = 28 days | Screen (-28 days) | On<br>Treatment <sup>1</sup> | At CMV reactivation <sup>2</sup> | AE follow<br>up <sup>3</sup> |
|---|---|---|---|---|
| REQUIRED ASSESSMENTS | | | | |
| Review of eligibility criteria, informed consent | Х | | | |
| Medical history | X | | | |
| ECOG PS⁴ | X | | | |
| Physical exam, vital signs <sup>5</sup> | X | X | X | Χ |
| AEs, concomitant medications | X | X | X | Χ |
| Drug diary | | X | X | |
| Assessment of contraception method <sup>6</sup> | X | | | |
| CMV disease assessment <sup>7</sup> | | | X | X |
| LABORATORY ASSESSMENTS | | | | |
| Complete blood cell count with differential (CBC) | X | X | X | X |
| Comprehensive metabolic profile (CMP) <sup>8</sup> | X | X | X | Χ |
| Prothrombin time (INR) | Х | | | |
| Urine pregnancy test in WOCBP | Х | Х | Х | X |
| HIV, hepatitis B, and hepatitis C screen <sup>9</sup> | X | | | |

| CMV IgG <sup>10</sup> | X | | | |
|---|---|---|---|---|
| CMV viral load <sup>11</sup> (at least every other week, weekly preferred) | X | X | X | X |
| CORRELATIVE STUDIES (SPECIMEN CO | OLLECTION) | | | |
| CMV Genotyping | | | Χ | |

- 1. On study visits will occur every 28 days (+/- 7 days). Treatment with letermovir should be continued for 90 after the last dose of alemtuzumab
- 2. CMV reactivation defined as CMV DNA by real time polymerase chain reaction >500 IU/mL
- 3. AE follow up to occur 30 days (+/- 7 days) from last dose of letermovir therapy. If patients have any ongoing toxicity related to letermovir, investigator should continue to monitor and provide appropriate supportive care. If patient has active CMV infection or reactivation, investigator should continue to monitor and provide appropriate treatment including antiviral therapy.
- 4. See Appendix 12.2
- 5. Vital signs include height, weight, blood pressure, heart rate, respiratory rate, temperature
- 6. See section 3.1 for acceptable methods of contraception
- 7. CMV disease assessment is a focused history and physical exam guided by known manifestations of CMV disease (see Appendix 12.1). CMV disease assessment is to be performed if reactivation occurs as defined in Section 10.2.
- 8. CMP should include at least the following: sodium, potassium, chloride, creatinine, glucose, calcium, phosphorus, total bilirubin, AST, ALT, alkaline phosphatase, albumin.
- 9. Screening to be completed with: HIV antibody, hepatitis B surface antibody, hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody. If hepatitis B surface antigen or core antibody is positive, hepatitis B viral load quantification with PCR should be ordered; if hepatitis C antibody is positive, viral load quantification by PCR should be ordered.
- 10. CMV IgG seropositivity may be confirmed up to 1 year prior to starting letermovir.
- 11. CMV viral load testing by PCR will be completed <u>at least every other week</u> while on therapy with letermovir. Weekly monitoring is preferred but can be reduced to every 2 weeks at the investigator's discretion. Window for screening is within 2 weeks of first dose of letermovir.

# 477 6.2 Biospecimen Studies and Procedures

- The correlative studies will include genotyping to evaluate mutations in CMV terminase complex
- 479 genes (UL51, UL56, UL89) through Viracor.

# 480 6.3 Source and Timing of Biospecimen Collections

- Peripheral blood of approximately 10 ml in EDTA (lavender top) tube will be inverted to mix anti-
- coagulant and then kept at room temperature until transport to the OSU Leukemia Tissue Bank
- 483 (LTB). Plasma and PBMCs will be separated and cryopreserved by standard methods. Samples
- 484 will be labeled with the study time point, collection date and protocol number as well as study
- 485 participant number. Frozen plasma samples would be batch analyzed after the completion of
- 486 the study for CMV genotyping studies.

#### 487 **6.4 Storage of Biospecimens**

488 Samples will be stored in OSU LTB.

#### 489 7 CRITERIA FOR DISEASE EVALUATION

- 490 CMV reactivation is defined in section 10.2. CMV disease will be defined as in Disease
- 491 Definitions Working Group of the Cytomegalovirus Drug Development Forum [71] (Appendix
- 492 12.1).

493

494

#### 8 LETERMOVIR INFORMATION

#### 8.1 Letermovir Description and Mechanism of Action

- Letermovir inhibits the CMV DNA terminase complex (pUL51, pUL56, and pUL89) which is
- 496 required for viral DNA processing and packaging. Biochemical characterization and electron

microscopy demonstrated that letermovir affects the production of proper unit length genomes and interferes with virion maturation. Genotypic characterization of virus resistant to letermovir confirmed that letermovir targets the terminase complex.

The median EC50 value of letermovir against a collection of clinical CMV isolates in a cell-culture model of infection was 2.1 nM (range = 0.7 nM to 6.1 nM, n = 74). There was no significant difference in EC50 value by CMV gB genotype (gB1=29; gB2=27; gB3=11; and gB4=3). No antagonism of the antiviral activity was seen when letermovir was combined with CMV DNA polymerase inhibitors (cidofovir, foscarnet, or ganciclovir).

# 8.2 Clinical Pharmacology

Letermovir has a molecular formula of C29H28F4N4O4 and a molecular weight of 572.55. The chemical name for letermovir is (4S)-2-[8-Fluoro-2-[4-(3-methoxyphenyl)piperazin-1-yl]-3-[2-methoxy-5(trifluoromethyl)phenyl]-3,4-dihydroquinazolin-4-yl] acetic acid. Letermovir is very slightly soluble in water.

510 The chemical structure of letermovir is:

# 511512

513514

497

498

499

500

501 502

503

504

505

506

507

508 509

#### 8.3 Pharmacokinetics and Drug Metabolism

The pharmacokinetic properties of letermovir are displayed in Table 2.

Table 2: Absorption, Distribution, Metabolism, Elimination (ADME), and Pharmacokinetic

516 Properties of letermovir

| Pharmacokinetics in HSCT Recipients | |
|---|---|
| Treatment Regimen | Steady-state median (90% prediction interval) AUC (ng•hr/mL) of letermovir |
| 480 mg oral once daily, no cyclosporine | 34,400 (16,900, 73,700) |
| 480 mg IV once daily, no cyclosporine | 100,000 (65,300, 148,000) |
| 240 mg oral once daily, with cyclosporine | 60,800 (28,700, 122,000) |
| 240 mg IV once daily, with cyclosporine | 70,300 (46,200, 106,000) |
| Pharmacokinetics in Healthy Subjects | |

| | IND Apploved. Zel ebzeze |
|---|---|
| Treatment Regimen | Steady-state geometric mean AUC and Cmax of letermovir |
| 480 mg oral once daily | Cmax: 13,000 ng/mL |
| | AUC: 71,500 ng•hr/mL |
| Dose proportionality | Greater than proportional following single and multiple oral or IV doses of letermovir 240 mg and 480 mg |
| Accumulation ratio <sup>†</sup> | Cmax: 1.03 |
| | AUC: 1.22 |
| Time to steady-state | 9-10 days |
| Absorption | |
| Bioavailability | Healthy subjects administered letermovir without cyclosporine: 94% at an oral dose range of 240 mg to 480 mg |
| | HSCT recipients administered letermovir without cyclosporine: 35% with 480 mg oral once daily |
| | HSCT recipients administered letermovir with cyclosporine: 85% with 240 mg oral once daily |
| Median Tmax (hr) | 45 min to 2.25 hr |
| Effect of food (relative to fasting) ‡ | AUC: 99.63% [84.27% - 117.80%] |
| | Cmax: 129.82% [104.35% -161.50%] |
| Distribution | |
| Mean steady-state volume of distribution | 45.5 L following IV administration in HSCT recipients |
| % <i>In vitro</i> bound to human plasma proteins | 99% across the concentration range of 0.2 to 50 mg/L |
| <i>In vitro</i> blood-to plasma ratio | 0.56 across the concentration range of 0.1 to 10 mg/L |
| Metabolism | |
| <i>In vitr</i> o metabolism | UGT1A1/1A3 (minor) |
| Drug-related component in plasma | 97% unchanged parent |
| | No major metabolites detected in plasma |
| Elimination | |
| Route of elimination | Hepatic uptake (OATP1B1/3) |
| Mean terminal t <sub>1/2</sub> (hr) | 12 hrs after dosing of letermovir 480 mg IV once daily |
| % of dose excreted in feces§ | 93% |

| | • |
|---|---|
| % of dose excreted in urine§ | <2% |
| % of unchanged drug excreted in feces§ | 70% |

<sup>\*</sup> Values were obtained in studies of healthy subjects unless otherwise indicated.

<sup>‡</sup> Values refer to geometric mean ratio [fed/fasted] percentage and 90% confidence interval back transformed from linear mixed-effects model performed on natural log-transformed values. The meal administered was a standard high fat and high calorie meal (33 grams protein, 65 grams carbohydrates, 58 grams fat; 920 total calories).

§ Single oral administration of radiolabeled letermovir in mass balance study.

517

#### 518 Specific Populations

- 519 Pediatric Population
- 520 The pharmacokinetics of letermovir in patients less than 18 years of age have not been
- 521 evaluated.
- 522 Age, Gender, Race, and Weight
- Age (18 to 78 years), gender, race (White vs. non-White), and body weight (up to 100 kg) did
- not have a clinically significant effect on the pharmacokinetics of letermovir.
- 525 Renal Impairment
- 526 Letermovir AUC was approximately 1.9-and 1.4-fold higher in subjects with moderate (eGFR
- 527 greater than or equal to 30 to 59 mL/min/1.73m2) and severe (eGFR less than 30
- 528 mL/min/1.73m2) renal impairment, respectively, compared to healthy subjects.
- 529 Hydroxypropyl betadex present in the intravenous letermovir formulation is mainly eliminated by
- 530 glomerular filtration. Decreased elimination of hydroxypropyl betadex has been reported in the
- 531 literature in patients with severe renal impairment.
- 532 Hepatic Impairment
- 533 Letermovir AUC was approximately 1.6-and 3.8-fold higher in subjects with moderate (Child-
- Pugh Class B [CP-B], score of 7-9) and severe (Child-Pugh Class C [CP-C], score of 10-15)
- hepatic impairment, respectively, compared to healthy subjects.
- 536 Drug Interaction Studies
- 537 Drug interaction studies were performed in healthy subjects with letermovir and drugs likely to
- 538 be co-administered or drugs commonly used as probes for pharmacokinetic interactions (see

<sup>†</sup> Based on geometric mean data.

539 Table **3** and

540 Table 4). 541 In vitro results indicate that letermovir is a substrate of drug metabolizing enzymes CYP3A, 542 CYP2D6, UGT1A1, and UGT1A3, and transporters OATP1B1/3 and P-qp. Oxidative 543 metabolism is considered to be a minor elimination pathway based on in vivo human data. 544 Inhibitors of OATP1B1/3 may result in increases in letermovir plasma concentrations. Changes 545 in letermovir plasma concentrations due to inhibition of P-qp or UGTs are not anticipated to be 546 clinically relevant. 547 Based on in vitro studies, the metabolism of letermovir is not mediated by CYP1A2, CYP2A6, 548 CYP2B6, CYP2C8, CYP2C9, CYP2C18, CYP2C19, CYP2E1, CYP4A11, UGT1A4, UGT1A6, 549 UGT1A7, UGT1A8, UGT1A9, UGT1A10, UGT2B4, UGT2B7, UGT2B15, or UGT2B17. The 550 transport of letermovir is not mediated by OATP2B1, OCT1, OAT1, BCRP, or MRP2 in vitro. 551 Letermovir is a time-dependent inhibitor and inducer of CYP3A in vitro. Co-administration of 552 letermovir with midazolam resulted in increased exposure of midazolam, indicating that the net 553 effect of letermovir on CYP3A is moderate inhibition (see

554 Table 4). Based on these results, co-administration of letermovir with CYP3A substrates may 555

increase the plasma concentrations of the CYP3A substrates (see

Table **4**). Letermovir is a reversible inhibitor of CYP2C8 *in vitro*. When co-administered with letermovir, plasma concentrations of CYP2C8 substrates are predicted to be increased (see

558 Table 4). Co-administration of letermovir reduced the exposure of voriconazole, most likely due 559 to the induction of voriconazole elimination pathways, CYP2C9 and CYP2C19. Co-560 administration of letermovir with CYP2C9 and CYP2C19 substrates may decrease the plasma 561 concentrations of the CYP2C9 and CYP2C19 substrates (see Table 5). Letermovir is an inducer 562 of CYP2B6 in vitro; the clinical relevance is unknown. 563 Letermovir inhibited efflux transporters P-qp, breast cancer resistance protein (BCRP), bile salt 564 export pump (BSEP), multidrug resistance-associated protein 2 (MRP2), OAT3, and hepatic uptake transporter OATP1B1/3 in vitro. Co-administration of letermovir with substrates of 565 566 OATP1B1/3 transporters (e.g. atorvastatin, a known substrate of CYP3A, OATP1B1/3, and 567 potentially BCRP) may result in a clinically relevant increase in plasma concentrations of 568 OATP1B1/3 substrates (see Table 5). There were no clinically relevant changes in plasma 569 concentrations of digoxin, a P-gp substrate, or acyclovir, an OAT3 substrate, following co-570 administration with letermovir in clinical studies (see

Table 4). The effect of letermovir on BCRP, BSEP, and MRP2 substrates was not evaluated in

- 572 clinical studies; the clinical relevance is unknown.
- 573 Based on *in vitro* results letermovir is not an inhibitor of CYP1A2, CYP2A6, CYP2C9, CYP2C19,
- 574 CYP2D6, CYP2E1, UGT1A4, UGT1A6, UGT1A9, or UGT2B7 and is not an inducer of CYP1A2.
- Letermovir is not an inhibitor of MRP2, OATP2B1, BSEP, OCT1, OCT2, or OAT1 *in vitro*.

# Table 3: Drug Interactions: Changes in Pharmacokinetics of Letermovir in the Presence of Co-administered Drug

577 578

579

| | Letermovir<br>Regimen | Geometric Mean Ratio [90% CI] of<br>Letermovir PK with/without<br>Co-administered Drug<br>(No Effect=1.00) | | |
|---|---|---|---|---|
| Drug | | AUC | Cmax | C24hr* |
| Immunosuppressants | | | | |
| 00 mg single<br>dose PO | 240 mg<br>once daily<br>PO | 2.11<br>(1.97, 2.26) | 1.48<br>(1.33, 1.65) | 2.06<br>(1.81, 2.35) |
| 1 g single<br>dose PO | 480 mg<br>once daily<br>PO | 1.18<br>(1.04, 1.32) | 1.11<br>(0.93, 1.34) | 1.39<br>(1.12, 1.74) |
| 5 mg single<br>dose PO | 80 mg<br>twice daily<br>PO | 1.02<br>(0.97, 1.07) | 0.92<br>(0.84, 1.00) | 1.02<br>(0.93, 1.12) |
| Abbreviations: PO= oral * C12hr for tacrolimus | | | | |
| | 00 mg single<br>dose PO 1 g single<br>dose PO 5 mg single<br>dose PO oral | Drug Ints Oo mg single dose PO 1 g single dose PO 5 mg single dose PO 5 mg single dose PO oral | Regimen (I AUC AUC AUC AUC | dministered Drug Regimen (No Effect=1.00 AUC Aux Cmax Ints 240 mg once daily PO 2.11 (1.97, 2.26) 1.48 (1.33, 1.65) 1 g single dose PO 480 mg once daily PO 1.18 (1.04, 1.32) 1.11 (0.93, 1.34) 5 mg single dose PO 80 mg twice daily PO 1.02 (0.97, 1.07) 0.92 (0.84, 1.00) oral oral 0.97, 1.07) 0.84, 1.00) |

# Table 4: Drug Interactions: Changes in Pharmacokinetics for Co-administered Drug in the Presence of Letermovir

| Co-<br>administered<br>Drug | administered administered | | Geometric Mean Ratio<br>[90% CI] of Co-administered Drug PK<br>with/without Letermovir<br>(No Effect=1.00) | | |
|---|---|---|---|---|---|
| Drug | | | AUC | Cmax | C24hr* |
| CYP3A Substrat | es | | | | |
| midazolam | 1 mg single<br>dose IV | 240 mg once<br>daily PO | 1.47<br>(1.37, 1.58) | 1.05<br>(0.94, 1.17) | 2.74<br>(2.16, 3.49) |
| midazolam | 2 mg single<br>dose PO | 240 mg once<br>daily PO | 2.25<br>(2.04, 2.49) | 1.72<br>(1.54, 1.92) | Not available |
| P-gp Substrates | | | | | |
| digoxin | 0.5 mg single<br>dose PO | 240 mg twice<br>daily PO | 0.88<br>(0.80, 0.96) | 0.75<br>(0.63, 0.89) | 0.90<br>(0.84, 0.96) |
| Immunosuppres | sants | | | | |
| cyclosporine | 50 mg single<br>dose PO | 240 mg once<br>daily PO | 1.66<br>(1.51, 1.82) | 1.08<br>(0.97, 1.19) | 2.19<br>(1.80, 2.66) |
| mycophenolate<br>mofetil | 1 g single dose<br>PO | 480 mg once<br>daily PO | 1.08<br>(0.97, 1.20) | 0.96<br>(0.82, 1.12) | 1.04<br>(0.86, 1.27) |
| tacrolimus | 5 mg single<br>dose PO | 480 mg once<br>daily PO | 2.42<br>(2.04, 2.88) | 1.57<br>(1.32, 1.86) | 2.53<br>(2.12, 3.03) |
| sirolimus | 2 mg single<br>dose PO | 480 mg once<br>daily PO | 3.40<br>(3.01, 3.85) | 2.76<br>(2.48, 3.06) | 3.15<br>(2.80, 3.55) |
| Antifungals and Antivirals | | | | | |
| acyclovir | 400 mg single<br>dose PO | 480 mg once<br>daily PO | 1.02<br>(0.87, 1.2) | 0.82<br>(0.71, 0.93) | 1.13<br>(0.94, 1.36) |
| posaconazole | 300 mg single<br>dose PO | 480 mg once<br>daily PO | 0.98<br>(0.82, 1.17) | 1.11<br>(0.95, 1.29) | 1.10<br>(0.94, 1.30) |
| voriconazole | 200 mg twice<br>daily PO | 480 mg once<br>daily PO | 0.56<br>(0.51, 0.62) | 0.61<br>(0.53, 0.71) | 0.49<br>(0.42, 0.57) |
| HMG-CoA Reductase Inhibitors | | | | | |
| atorvastatin | 20 mg single<br>dose PO | 480 mg once<br>daily PO | 3.29<br>(2.84, 3.82) | 2.17<br>(1.76, 2.67) | 3.62<br>(2.87, 4.55) |
| Oral Contracept | ives | | | | |
| ethinyl estradiol<br>(EE) | 0.03 mg EE<br>single dose PO | 480 mg once<br>daily PO | 1.42<br>(1.32, 1.52) | 0.89<br>(0.83, 0.96) | 1.57<br>(1.45, 1.70) |
| /levonorgestrel<br>(LNG) | 0.15 mg LNG<br>single dose PO | | 1.36<br>(1.30, 1.43) | 0.95<br>(0.86, 1.04) | 1.38<br>(1.32, 1.46) |
| Abbreviations: PC * C12hr reported | | | | | |

581

Table 5: Potentially Significant Drug Interactions: Alteration in Dose May Be Recommended Based on Results from Drug Interaction Studies or Predicted Interactions\* (Information in the Table Applies to Co-administration of Letermovir and the Concomitant Drug without Cyclosporine, Unless Otherwise Indicated)

584

585

586

| Concomitant Drug<br>Class and/or Clearance<br>Pathway: Drug Name | Effect on<br>Concentration <sup>†</sup> | Clinical Comments |
|---|---|---|
| Anti-arrhythmic agents | | |
| amiodarone | ↑ amiodarone | Close clinical monitoring for adverse events related to amiodarone is recommended during coadministration. Frequently monitor amiodarone concentrations when amiodarone is coadministered with letermovir. |
| Anticoagulants | | |
| warfarin | ↓ warfarin | When letermovir is co-administered with warfarin, frequently monitor International Normalized Ratio (INR)§. |
| Anticonvulsants | | |
| phenytoin | ↓ phenytoin | When letermovir is co-administered with phenytoin, frequently monitor phenytoin concentrations§. |
| Antidiabetic agents | | |
| Examples: glyburide, repaglinide, rosiglitazone | glyburide, repaglinide | When letermovir is co-administered with glyburide, repaglinide, or rosiglitazone, frequently monitor glucose concentrations§. |
| Tosigitazone | ↑ rosiglitazone | When letermovir is co-administered with cyclosporine, use of repaglinide is not recommended. |
| Antifungals | | |
| voriconazole <sup>‡</sup> | ↓ voriconazole | If concomitant administration of voriconazole is necessary, closely monitor for reduced effectiveness of voriconazole§. |
| Antimycobacterial | | |
| rifampin | ↓ letermovir | Co-administration of letermovir and rifampin is not recommended. |
| Antipsychotics | | |

| pimozide | ↑ pimozide | Co-administration is <b>contraindicated</b> due to risk of QT prolongation and torsades de pointes |
|---|---|---|
| Ergot alkaloids | Ergot alkaloids | |
| ergotamine,<br>dihydroergotamine | ↑ ergotamine,<br>dihydroergotamine | Co-administration is <b>contraindicated</b> due to risk of ergotism |
| HMG-CoA Reductase Inh | ibitors | , |
| atorvastatin <sup>‡</sup> | ↑ atorvastatin | When letermovir is co-administered with atorvastatin, do not exceed an atorvastatin dosage of 20 mg daily§. Closely monitor patients for myopathy and rhabdomyolysis. |
| | | When letermovir is co-administered with cyclosporine, use of atorvastatin is not recommended. |
| pitavastatin,<br>simvastatin | ↑ HMG-CoA<br>reductase inhibitors | Co-administration of letermovir and pitavastatin or simvastatin is not recommended. |
| | | When letermovir is co-administered with cyclosporine, use of either pitavastatin or simvastatin is contraindicated due to significantly increased pitavastatin or simvastatin concentrations and risk of myopathy or rhabdomyolysis |
| fluvastatin, lovastatin,<br>pravastatin, rosuvastatin | ↑ HMG-CoA<br>reductase inhibitors | When letermovir is co-administered with these statins, a statin dosage reduction may be necessary§. Closely monitor patients for myopathy and rhabdomyolysis. |
| | | When letermovir is co-administered with cyclosporine, use of lovastatin is not recommended. |
| | | When letermovir is co-administered with cyclosporine, refer to the statin prescribing information for specific statin dosing recommendations. |
| Immunosuppressants | | |
| | ↑ cyclosporine<br>↑ letermovir | Decrease the dosage of letermovir to 240 mg once daily |
| | | Frequently monitor cyclosporine whole blood concentrations during treatment and after discontinuation of letermovir and adjust the dose of cyclosporine accordingly§. |

| | | · |
|---|---|---|
| sirolimus <sup>‡</sup> | ↑ sirolimus | When letermovir is co-administered with sirolimus, frequently monitor sirolimus whole blood concentrations during treatment and after discontinuation of letermovir and adjust the dose of sirolimus accordingly§. |
| | | When letermovir is co-administered with cyclosporine and sirolimus, refer to the sirolimus prescribing information for specific sirolimus dosing recommendations§. |
| tacrolimus‡ | ↑ tacrolimus | Frequently monitor tacrolimus whole blood concentrations during treatment and after discontinuation of letermovir and adjust the dose of tacrolimus accordingly§. |
| Proton pump inhibitors | | |
| omeprazole | ↓omeprazole | Clinical monitoring and dose adjustment may be needed. |
| pantoprazole | ↓ pantoprazole | Clinical monitoring and dose adjustment may be needed. |
| CYP3A Substrates | | |
| Examples: alfentanil, fentanyl, midazolam, and quinidine | ↑ CYP3A substrate | When letermovir is co-administered with a CYP3A substrate, refer to the prescribing information for dosing of the CYP3A substrate with a moderate CYP3A inhibitor§. |
| | | When letermovir is co-administered with cyclosporine, the combined effect on CYP3A substrates may be similar to a strong CYP3A inhibitor. Refer to the prescribing information for dosing of the CYP3A substrate with a strong CYP3A inhibitor§. |
| | | CYP3A substrates pimozide and ergot alkaloids are contraindicated |

<sup>\*</sup> This table is not all inclusive.

588

589

591

592

593

594

# 8.4 Preparation, Storage, and Administration: Oral Formulation

590 Letermovir tablets are supplied in two formulations:

- Letermovir 240 mg tablet: yellow oval tablet with "591" on one side and Merck logo on the other side.
- Letermovir 480 mg tablet: pink oval, bi-convex tablet with "595" on one side and Merck logo on the other side.

<sup>&</sup>lt;sup>†</sup> ↓ =decrease, ↑=increase

<sup>&</sup>lt;sup>‡</sup>These interactions have been studied [see Package Insert: Clinical Pharmacology (12.3)].

<sup>§</sup> Refer to the respective prescribing information.

- Letermovir tablets contain either 240 mg or 480 mg of letermovir and the following inactive
- 596 ingredients: colloidal silicon dioxide, croscarmellose sodium, magnesium stearate,
- 597 microcrystalline cellulose, povidone 25, and film-coated with a coating material containing the
- following inactive ingredients: hypromellose 2910, iron oxide red (only for 480 mg tablets), iron
- oxide yellow, lactose monohydrate, titanium dioxide, and triacetin, Carnauba wax is added as a
- 600 polishing agent.
- Tablets should be swallowed whole with or without food.
- Store letermovir tablets in the original package until use.
- Store letermovir tablets at 20°C to 25°C (68°F to 77°F); excursions permitted to 15°C to 30°C
- 604 (59°F to 86°F)

# 8.5 Preparation, Storage, and Administration: Intravenous formulation

- 606 Letermovir injection is supplied in 30 mL single-dose vials containing either 240 mg/12 mL per
- or 480 mg/24 mL per vial (20 mg/mL). The preparation and administration
- instructions are the same for either dose.
- 609 Letermovir vials are for single use only. Discard any unused portion.
- 610 Preparation and Administration Instructions
- Letermovir must be diluted prior to intravenous (IV) use.
- Inspect vial contents for discoloration and particulate matter prior to dilution. Letermovir injection is a clear colorless solution. Do not use the vial if the solution is discolored or contains visible particles.
- Do not shake letermovir vial.
- Add one single-dose vial of letermovir injection into a 250 mL pre-filled IV bag containing either 0.9% Sodium Chloride Injection, USP or 5% Dextrose Injection, USP and mix bag gently. Do not shake. Only 0.9% Sodium Chloride and 5% Dextrose are chemically and physically compatible with letermovir injection.
  - Use compatible IV bags and infusion set materials. Letermovir injection is compatible with the following IV bags and infusion set materials. Letermovir injection is not recommended with any IV bags or infusion set materials not listed below (note that letermovir injection is not recommended for use with polyurethane-containing IV administration set tubing).
- 624 IV Bags Materials:

620

621

622

- Polyvinyl chloride (PVC), ethylene vinyl acetate (EVA) and polyolefin (polypropylene and polyethylene)
- 627 <u>Infusion Sets Materials:</u>
- PVC, polyethylene (PE), polybutadiene (PBD), silicone rubber (SR), styrene-butadiene
- 629 copolymer (SBC), styrene-butadiene-styrene copolymer (SBS), polystyrene (PS)
- 630 Plasticizers:

Diethylhexyl phthalate (DEHP), tris (2-ethylhexyl) trimellitate (TOTM), benzyl butyl phthalate (BBP)

## 633 <u>Catheters:</u>

635

636

637

638

639

640

641

642

643

644

645

646

654

655

656

657

658

659

660

661

662

663

664

665

Radiopaque polyurethane

- Once diluted, the solution of letermovir is clear, and ranges from colorless to yellow.
   Variations of color within this range do not affect the quality of the product. Parenteral drug products should be inspected visually for particulate matter and discoloration prior to administration, whenever solution and container permit. Discard if discoloration or visible particles are observed.
- The diluted solution is stable for up to 24 hours at room temperature or up to 48 hours under refrigeration at 2°C to 8°C (36°F to 46°F) (this time includes storage of the diluted solution in the intravenous bag through the duration of infusion).
- Administer the entire contents of the intravenous bag by intravenous infusion via a
  peripheral catheter or central venous line at a constant rate over 1 hour. Do not
  administer as an IV bolus injection.

#### Compatible Drug Products:

The physical compatibility of letermovir injection with selected injectable drug products was evaluated in two commonly available diluents. Letermovir should not be co-administered through the same intravenous line (or cannula) with other drug products and diluent combinations except those listed below. Refer to the respective prescribing information of the co-administered drug(s) to confirm compatibility of simultaneous co-administration.

652 List of Compatible Drug Products when letermovir and Drug Products are Prepared in 0.9% 653 Sodium Chloride Injection, USP:

Ampicillin sodium, ampicillin sodium/sulbactam sodium, anti-thymocyte globulin, caspofungin, daptomycin, fentanyl citrate, fluconazole, furosemide, human insulin, magnesium sulfate, methotrexate, micafungin.

List of Compatible Drug Products when letermovir and Drug Products are Prepared in 5% Dextrose Injection, USP:

Amphotericin B (lipid complex)\*, anidulafungin, cefazolin sodium, ceftaroline, ceftriaxone sodium, doripenem, famotidine, folic acid, ganciclovir sodium, hydrocortisone sodium succinate, morphine sulfate, norepinephrine bitartrate, pantoprazole sodium, potassium chloride, potassium phosphate, tacrolimus, telavancin, tigecycline.

\*Amphotericin B (lipid complex) is compatible with letermovir. However, Amphotericin B (liposomal) is incompatible (see below)

#### Incompatible Drug Products

Letermovir injection is physically incompatible with amiodarone hydrochloride, amphotericin B (liposomal), aztreonam, cefepime hydrochloride, ciprofloxacin, cyclosporine, diltiazem hydrochloride, filgrastim, gentamicin sulfate, levofloxacin, linezolid, lorazepam, midazolam HCl, mycophenolate mofetil hydrochloride, ondansetron, palonosetron.

- 670 Storage
- Store letermovir injection vials at 20°C to 25°C (68°F to 77°F); excursions permitted to 15°C to
- 672 30°C (59°F to 86°F).
- Store in the original carton to protect from exposure to light.
- 674 8.6 Non Clinical Toxicology
- 8.6.1 Carcinogenesis, Mutagenesis, Impairment of Fertility
- 676 Carcinogenesis and Mutagenesis
- 677 Letermovir was not genotoxic in *in vitro* or *in vivo* assays, including microbial mutagenesis
- 678 assays, chromosomal aberration in Chinese hamster ovary cells, and in an in vivo mouse
- 679 micronucleus study.
- 680 Carcinogenicity studies with letermovir have not been conducted.
- 681 Impairment of Fertility
- In a fertility and early embryonic development study in rats, no effects of letermovir on female
- 683 fertility were observed at letermovir exposures (AUC) approximately 5 times higher than human
- exposure at the RHD.
- In male rat fertility studies, decreased fertility associated with irreversible testicular toxicity was
- 686 observed at
- 687 ≥180 mg/kg/day (greater than or equal to 3 times the human exposure at the RHD). No fertility
- or testicular effects were observed at dose levels resulting in letermovir exposures (AUC) similar
- to human exposure at the RHD [see Nonclinical Toxicology (13.2)].
- 690 8.6.2 Animal Toxicology and Pharmacology
- 691 Testicular toxicity in rats observed at ≥180 mg/kg/day (greater than or equal to 3 times the
- 692 human exposure at the RHD) was characterized by decreased testis weight, bilateral
- seminiferous tubular degeneration, decreased sperm count and motility, and resultant
- decreased male fertility. Male reproductive system toxicities were not observed in either a
- 695 monkey testicular toxicity study up to 240 mg/kg/day (approximately 2 times higher than human
- 696 exposure at the RHD), or a general toxicology study in mice up to 250 mg/kg/day
- 697 (approximately 3 times higher than human exposure at the RHD).
- 698 8.7 Clinical Studies
- To evaluate letermovir prophylaxis as a preventive strategy for CMV infection or disease in
- transplant recipients at high risk for CMV reactivation, the efficacy of letermovir was assessed in
- 701 a multicenter, double-blind, placebo-controlled Phase 3 Trial (P001, NCT02137772) in adult
- 702 CMV-seropositive recipients [R+] of an allogeneic hematopoietic stem cell transplant (HSCT).
- 703 Subjects were randomized (2:1) to receive either letermovir at a dose of 480 mg once daily
- adjusted to 240 mg when co-administered with cyclosporine, or placebo. Randomization was
- stratified by investigational site and risk level for CMV reactivation at the time of study entry.
- 706 Study drug was initiated after HSCT (at any time from Day 0 to Day 28 post-transplant) and
- 707 continued through Week 14 post-transplant. Study drug was administered either orally or
- intravenously; the dose of letermovir was the same regardless of the route of administration.
- 709 Subjects received CMV DNA monitoring weekly until post-transplant Week 14 and then bi-
- 710 weekly until post- transplant Week 24, with initiation of standard-of-care CMV pre-emptive
- 711 therapy if CMV viremia was considered clinically significant. Subjects had continued follow-up
- 712 through Week 48 post-transplant.
- Among the 565 treated subjects, 70 subjects were found to have CMV viremia prior to study
- drug initiation and were therefore excluded from the efficacy analyses. The efficacy population
- 715 consisted of 325 subjects who received letermovir (including 91 subjects who received at least
- one IV dose) and 170 who received placebo (including 41 subjects who received at least one IV
- 717 dose). The IV formulation of letermovir was used at investigators' discretion in subjects who
- 718 were unable to take oral therapy (e.g., unable to tolerate oral intake). The median time to
- starting study drug was 8 days after transplantation. Thirty-four percent (34%) of subjects were
- engrafted at baseline. The median age was 55 years (range: 18 to 76 years); 57% were male;
- 721 84% were White; 9% were Asian; 2% were Black or African American; and 7% were Hispanic or
- 722 Latino.
- 723 At baseline, 30% of all subjects had one or more of the following factors associated with
- 724 increased risk for CMV reactivation (high risk stratum): Human Leukocyte Antigen (HLA)-related
- donor with at least one mismatch at one of the following three HLA-gene loci: HLA-A, -B or –DR;
- haploidentical donor; unrelated donor with at least one mismatch at one of the following four
- 727 HLA-gene loci: HLA-A, -B, -C and -DRB1; use of umbilical cord blood as stem cell source; use
- of ex vivo T-cell-depleted grafts; Grade 2 or greater Graft- Versus-Host Disease (GVHD)
- 729 requiring systemic corticosteroids. The remaining 70% of subjects did not meet any of these
- high risk stratum criteria and were therefore included in the low risk stratum. Additionally, 48%
- of subjects received a myeloablative regimen, 51% were receiving cyclosporine, and 43% were
- 732 receiving tacrolimus. The most common primary reasons for transplant were acute myeloid
- 733 leukemia (38%), myelodysplastic syndrome (16%), and lymphoma (12%).
- 734 Clinically Significant CMV Infection
- 735 The primary efficacy endpoint of Trial P001 was the incidence of clinically significant CMV
- 736 infection through Week 24 post-transplant (prophylaxis failure). Clinically significant CMV
- 737 infection was defined as the occurrence of either CMV end-organ disease, or initiation of anti-
- 738 CMV pre-emptive therapy (PET) based on documented CMV viremia (using the Roche
- 739 COBAS® AmpliPrep/COBAS TaqMan® assay, LLoQ is 137 IU/mL, which is approximately 150
- 740 copies/mL) and the clinical condition of the subject. The protocol-
- specified guidance for CMV DNA thresholds for the initiation of PET during the treatment period
- 742 was ≥ 150 copies/mL or > 300 copies/mL for subjects in the high and low risk strata,
- 743 respectively. From Week 14 through Week 24, the threshold was >300 copies/mL for both high
- and low risk strata subjects. The Non- Completer=Failure (NC=F) approach was used, where
- subjects who discontinued from the trial prior to Week 24 post-transplant or had a missing
- outcome at Week 24 post-transplant were counted as failures.
- 747 Efficacy results from Trial P001 are shown in .

748 **Table 6**.

# Table 6: Trial P001 Efficacy Results in HSCT Recipients (NC=F Approach, FAS Population) Through Week 24

| Parameter | Letermovir<br>(N=325) | Placebo<br>(N=170) |
|---|---|---|
| Proportion of subjects who failed prophylaxis Reasons for failures* | 38% | 61% |
| Clinically significant CMV infection by Week 24 <sup>†</sup> | 18% | 42% |
| Initiation of PET based on documented CMV viremia | 16% | 40% |
| CMV end-organ disease | 2% | 2% |
| Discontinued from study before Week 24‡ | 17% | 16% |
| Missing outcome in Week 24 visit window | 3% | 3% |
| Stratum-adjusted treatment difference (Letermovir-Placebo)§ | | |
| Difference (95% CI) | -23.5 (-32.5, -14.6)¶ | |

<sup>\*</sup> The categories of failure are mutually exclusive and based on the hierarchy of categories in the order listed.

Note: FAS=Full analysis set; FAS includes randomized subjects who received at least one dose of study medication, and excludes subjects with detectable CMV DNA at baseline. Approach to handling missing values: Non-Completer=Failure (NC=F) approach. With NC=F approach, failure was defined as all subjects who developed clinically significant CMV infection or prematurely discontinued from the study or had a missing outcome through Week 24 post-transplant visit window.

751752

753

749 750

Efficacy results were consistent across high and low risk strata for CMV reactivation. The time to clinically significant CMV infection is shown in

<sup>&</sup>lt;sup>†</sup>Through Week 14, 8% of subjects in the letermovir group and 39% of subjects in the placebo group experienced clinically significant CMV infection.

<sup>‡</sup> Reasons for discontinuation included adverse event, death, lost to follow-up, physician decision, and withdrawal by subject.

<sup>§ 95%</sup> CI and p-value for the treatment differences in percent response were calculated using stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of sample size per arm for each stratum (high or low risk).

<sup>¶</sup>p-value <0.0001.

754 Figure **1**.

755

Figure 1: P001: Kaplan-Meier Plot of Time to Onset of Clinically Significant CMV Infection Through Week 24 Post-Transplant in HSCT Recipients (FAS Population)



| Number of Subj | ects at Risk | | |
|----------------|--------------|-----|-----|
| — Letermovir | 325 | 270 | 212 |
| Placebo | 170 | 85 | 70 |

Post-hoc analysis demonstrated that among letermovir-treated subjects, inclusion in the high risk stratum for CMV reactivation at baseline, occurrence of GVHD, and steroid use at any time after randomization may be associated with the development of clinically significant CMV infection between Week 14 and Week 24 post-transplant.

#### 763 Mortality

The Kaplan-Meier event rate for all-cause mortality in the letermovir vs. placebo groups was 12% vs. 17% at Week 24 post-transplant, and 24% vs. 28% at Week 48 post-transplant.

#### 8.8 Adverse Events

#### Adult CMV-seropositive Recipients [R+] of an Allogeneic HSCT

The safety of letermovir was evaluated in one Phase 3 randomized, double-blind, placebo-controlled trial (P001) in which 565 subjects were randomized and treated with letermovir (N=373) or placebo (N=192) through Week 14 post-transplant. Adverse events were those reported while subjects were on study medication or within two weeks of study medication completion/discontinuation. The mean time for reporting adverse events and laboratory abnormalities was approximately 22% longer in the letermovir arm compared to the placebo arm.

#### 775 Cardiac Adverse Events:

776 The cardiac adverse event rate (regardless of investigator-assessed causality) was higher in 777 subjects receiving letermovir (13%) compared to subjects receiving placebo (6%). The most 778 common cardiac adverse events were tachycardia (reported in 4% of letermovir subjects and in 779 2% of placebo subjects) and atrial fibrillation (reported in 3% of letermovir subjects and in 1% of 780 placebo subjects). Among those subjects who experienced one or more cardiac adverse events, 781 85% of letermovir and 92% of placebo subjects had events reported as mild or moderate in 782 severity.

#### Common Adverse Events

783

787

788

789

790

791

792

793

794

795

798

784 The rate of adverse events occurring in at least 10% of subjects in the letermovir group and at a 785 frequency at least 2% greater than placebo are outlined in Table 7.

786 Table 7: Trial P001 All Grade Adverse Events Reported in ≥ 10% of Letermovir-Treated HSCT Recipients at a Frequency at least 2% Greater than Placebo

| Adverse Events | Letermovir<br>(N=373) | Placebo<br>(N=192) |
|------------------|-----------------------|--------------------|
| nausea | 27% | 23% |
| diarrhea | 26% | 24% |
| vomiting | 19% | 14% |
| peripheral edema | 14% | 9% |
| cough | 14% | 10% |
| headache | 14% | 9% |
| fatigue | 13% | 11% |
| abdominal pain | 12% | 9% |

Overall, similar proportions of subjects in each group discontinued study medication due to an adverse event (13% of letermovir subjects vs. 12% of placebo subjects). The most frequently reported adverse event that led to study drug discontinuation was nausea, occurring in 2% of letermovir subjects and 1% of placebo subjects. Hypersensitivity reaction, with associated moderate dyspnea, occurred in one subject following the first infusion of IV letermovir after switching from oral letermovir, leading to treatment discontinuation.

#### **Laboratory Abnormalities**

796 Selected laboratory abnormalities reported during treatment or within 2 weeks of stopping 797 treatment are presented in Table 8.

**Table 8: Trial P001 Selected Laboratory Abnormalities** 

| | Letermovir<br>N=373 | Placebo<br>N=192 |
|---|---|---|
| Absolute neutrophil count (cells/µL) | | |
| < 500 | 19% | 19% |

| 500 – < 750 | 4% | 7% |
|--------------------------|-----|-----|
| 750 – < 1000 | 8% | 9% |
| Hemoglobin (g/dL) | | |
| < 6.5 | 2% | 1% |
| 6.5 – < 8.0 | 14% | 15% |
| 8.0 – < 9.5 | 41% | 43% |
| Platelets (cells/µL) | | |
| < 25000 | 27% | 21% |
| 25000 - < 50000 | 17% | 18% |
| 50000 - < 100000 | 20% | 30% |
| Serum creatinine (mg/dL) | | |
| > 2.5 | 2% | 3% |
| > 1.5 – 2.5 | 17% | 20% |

799 800

801

802

803

804

The median time to engraftment (defined as absolute neutrophil count ≥ 500/mm3 on 3 consecutive days after transplantation) was 19 days in the letermovir group and 18 days in the placebo group.

#### 9 REGULATORY AND REPORTING REQUIREMENTS

#### 9.1 Adverse Events (AEs)

Definition: any unfavorable medical occurrence in a human subject including any abnormal sign, symptom, or disease.

For the purposes if this study, "Adverse Event" or "AE" shall mean any untoward medical occurrence iin a Study subject who is administered the Study Drug (letermovir) regardless of whether or not a causal relationship with the Study Drug exists. By way of example and without limitation, an AE can be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of

the Study Drug.

Grading: the descriptions and grading scales found in the revised NCI Common Terminology
Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting. A copy
of the CTCAE version 5.0 can be downloaded from the CTEP website.

Attribution (relatedness), Expectedness, and Seriousness: the definitions for the terms listed that should be used are those provided by the Department of Health and Human Services'

Office for Human Research Protections (OHRP). A copy of this guidance can be found on

819 OHRP's website:

820 http://www.hhs.gov/ohrp/policy/advevntguid.html

#### 821 Unanticipated Problems Definition:

822

823

824

825

826

827

828

829

830

831

853

- unexpected (in terms of nature, severity, or frequency) given (a) the research procedures
  that are described in the protocol-related documents, such as the IRB- approved
  research protocol and informed consent document; and (b) the characteristics of the
  subject population being studied;
- related or possibly related to participation in the research ("possibly related" means there
  is a reasonable possibility that the incident, experience, or outcome may have been
  caused by the procedures involved in the research);
  - Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

## 832 9.2 Serious Adverse Events (SAEs)

- "Serious Adverse Event" or "SAE" shall mean any untoward medical occurrence in a Study subject who is administered the Study Drug (letermovir) which meets one or more of the seriousness criteria outlined below.
- An adverse event should be classified as a serious adverse event if the following seriousness criteria are met:
- It results in death (i.e., the adverse event actually causes or leads to death)
- It is life threatening (i.e., the adverse event, in the view of the investigator, places the subject at immediate risk of death. It does not include an adverse event that, had it occurred in a more severe form, might have caused death.).
- It requires or prolongs inpatient hospitalization.
- It results in persistent or significant disability/incapacity (i.e., the adverse event results in substantial disruption of the subject's ability to conduct normal life functions).
- It results in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the IMP.
- It is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the subject or may require medical/surgical intervention to prevent one of the outcomes listed above).
- "Suspected Unexpected Serious Adverse Reaction" or "SUSAR" shall mean any Serious
   Adverse Event, the nature, severity or frequency of which is not consistent with information in
   the most current Summary of Product Characteristics (SPC) or Package Insert.

#### 9.3 Noncompliance

Definition: failure to follow any applicable regulation or institutional policies that govern human subjects research or failure to follow the determinations of the IRB. Noncompliance may occur due to lack of knowledge or due to deliberate choice to ignore regulations, institutional policies, or determinations of the IRB.

#### 858 9.4 Serious Noncompliance

Definition: noncompliance that materially increases risks, that results in substantial harm to subjects or others, or that materially compromises the rights or welfare of participants.

#### 861 9.5 Reporting to the OSU IRB

- The OSU PI is required to promptly notify the IRB of the following events:
- Any unanticipated problems involving risks to participants or others which occur at OSU, or that impacts participants or the conduct of the study.
- Noncompliance with federal regulations or the requirements or determinations of the IRB.
- Receipt of new information that may impact the willingness of participants to participate or continue participation in the research study.
- These events must be reported to the IRB within the time frames outlined in the IRB policy.

### 869 9.6 Reporting to the sponsor

- Principal investigator shall forward to Merck's Global Pharmacovigilance ("Merck GPV") group,
- any SAE or SUSAR, including, but not limited to, all initial and follow up information involving
- any study subject in the study. Notification shall be in the form of a completed CIOMS
- 873 I/MedWatch (or other mutually agreed upon format) within two (2) business days of but not
- longer than three (3) calendar days of receipt of this information. This information shall be
- 875 transmitted to Merck GPV using the contact information provided below or such other modified
- 876 contact information as provided by Merck in writing. All information shall be transmitted in the
- 877 English language and contain the reporter's name and the study subject identifier code. SUSAR
- information will be reported unblinded if the study drug has been blinded in the study.
- 879 Randomization codes for all other SAEs will be provided to Merck GPV at end of study if the
- 880 Study Drug has been blinded in the study.
- 881 SAE reports and any other relevant safety information are to be forwarded to Merck GPV
- 882 facsimile number: 215-661-6229.

883

888

889

890

891

892

893

894

#### 9.7 Reporting to the FDA

- The conduct of the study will comply with all FDA safety reporting requirements. **PLEASE**
- 885 NOTE THAT REPORTING REQUIREMENTS FOR THE FDA DIFFER FROM REPORTING
- 886 **REQUIREMENTS FOR THE IRB.** It is the responsibility of the investigator to report any
- 887 unanticipated problem to the FDA as follows:
  - Report any unexpected fatal or life-threatening adverse experiences associated with use
    of the drug (i.e., there is a reasonable possibility that the experience may have been
    caused by the drug) by telephone or fax no later than 7 calendar days after initial receipt
    of the information. A life-threatening adverse experience is defined as any adverse drug
    experience that places the subject (in the view of the investigator) at immediate risk of
    death from the reaction as it occurred, i.e., it does not include a reaction that, had it
    occurred in a more severe form, might have caused death.

895 Report any serious, unexpected adverse experiences, as well as results from animal 896 studies that suggest significant clinical risk within 15 calendar days after initial receipt of 897 this information. A serious adverse drug experience is defined as any adverse drug 898 experience occurring at any dose that results in any of the following outcomes: 899 o Death 900 A life-threatening adverse drug experience 901 Inpatient hospitalization or prolongation of existing hospitalization 902 o A persistent or significant disability/incapacity (i.e., a substantial disruption of a 903 person's ability to conduct normal life functions) 904 A congenital anomaly/birth defect 905 o Any other experience which, based upon appropriate medical judgment, may 906 jeopardize the subject and may require medical or surgical intervention to 907 prevent one of the outcomes listed above 908 An unexpected adverse drug experience is defined as any adverse drug experience, the 909 specificity or severity of which is not consistent with the current investigator brochure (or risk 910 information, if an IB is not required or available). 911 All MedWatch forms will be sent by the investigator or investigator's team to the FDA (refer to 912 the FDA website to obtain the current address and fax number for the Center for Drug 913 Evaluation and Research Division of Oncology Drug Products).

#### 914 9.8 Timeframe for Reporting Required Events

915 Reportable adverse events will be tracked for 30 days following the last day of study treatment.

| Deaths | |
|---|---|
| Any reportable death while on study or within 30 days of study | Immediately, within 24 hours, to PI and the IRB |
| Any reportable death while off study | Immediately, within 24 hours, to PI and the IRB |
| Adverse Events/Unanticipated Problems | |
| Any reportable adverse events as described in Sections 9.1 and 9.2 (other than death) and 9.9 | Immediately, within 24 hours to PI and within required time frame to the IRB (per local policy) and within 7 or 15 calendar days to the FDA |
| All adverse events regardless of grade and attribution should be submitted cumulatively | Include in DSM report |
| Noncompliance and Serious Noncompliance | |

| All noncompliance and serious | Immediately, within 24 hours, to PI and |
|---|---|
| noncompliance as described in Sections 9.3 | within required time frame to the IRB (per |
| and 9.4 | local policy) |

916

917

#### 9.9 Overdose

- In this trial, an overdose is any dose higher than two times the dose specified in section 4.
- 919 If an adverse event(s) is associated with ("results from") the overdose of Sponsor's product, the
- 920 adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria
- are met. If a dose of Sponsor's product meeting the protocol definition of overdose is taken
- 922 without any associated clinical symptoms or abnormal laboratory results, the overdose is
- 923 reported as a non-serious Event of Clinical Interest (ECI), using the terminology "accidental or
- 924 intentional overdose without adverse effect." All reports of overdose with and without an adverse
- event must be reported within 24 hours to the Sponsor either by electronic media or paper.
- 926 There is no specific antidote for overdose with letermovir. In case of overdose, it is
- 927 recommended that the patient be monitored for adverse reactions and appropriate symptomatic
- 928 treatment be instituted.

929

930

932

943

- It is unknown whether dialysis will result in meaningful removal of letermovir from systemic
- 931 circulation.

## 9.10 Pregnancies

- 933 Pregnancies and suspected pregnancies (including a positive pregnancy test regardless of age
- or disease state) of a woman occurring while on study or within 28 days of her last dose of study
- 935 drug are considered immediately reportable events. Protocol therapy is to be discontinued
- 936 immediately. The pregnancy, suspected pregnancy, or positive pregnancy test must be reported
- 937 within 24 hours.
- 938 All subjects who become pregnant must be followed to the completion/termination of the
- 939 pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform
- 940 mole, blighted ovum, fetal death, intrauterine death, miscarriage and stillbirth must be reported
- 941 as serious events (Important Medical Events). CRFs will be used to report pregnancies and
- 942 pregnancy outcomes.

#### 9.11 Data and safety monitoring

- The data and safety monitoring plan will involve the continuous evaluation of safety, data quality
- and data timeliness. Investigators will conduct continuous review of data and patient safety at
- the regular protocol review meeting at least monthly. The PI of the trial will review toxicities and
- responses of the trial where applicable and determine if the risk/benefit ratio of the trial changes.
- 948 Frequency and severity of adverse events will be reviewed by the PI and compared to what is
- 849 known about the agent/device from other sources; including published literature, scientific
- 950 meetings and discussions with sponsors, to determine if the trial should be terminated before
- completion. Serious adverse events and responses will also be reviewed by the OSUCCC Data

- and Safety Monitoring Committee (DSMC). The PI will also submit a progress report that will be
- 953 reviewed by the committee per the DSMC plan. All reportable Serious Adverse Events (SAE)
- will be reported to the IRB of record as per the policies of the IRB.

#### 955 **9.11.1 Data Submission**

- 956 The study will be managed per OSU Clinical Trial Office. Data will be directly entered into the
- 957 OSU OnCore database.

#### 958 **9.11.2 Auditing**

- 959 As the study sponsor, The Ohio State University Comprehensive Cancer Center (OSUCCC) will
- audit the trial per OSU policies. Audits will be performed by the OSUCCC Clinical Research
- 961 Audit Team.

962

#### 9.12 Ethical Considerations

- The study will be conducted in accordance with ethical principles founded in the Declaration of
- 964 Helsinki. Investigators and study staff will undergo training on Good Clinical Practice (GCP)
- 965 through the Collaborative Institutional Training Initiative (CITI). GCP training sets the standard
- 966 for the design, conduct, recording, and reporting of studies involving human subjects, ensuring
- that study subjects rights, safety, and well-being are protected. The IRB will review all
- 968 appropriate study documentation in order to safeguard the rights, safety and wellbeing of the
- patients. The study will only be conducted at sites where IRB approval has been obtained. The
- protocol, informed consent form, written information given to the patients (including pill diaries),
- 971 safety updates, annual progress reports, and any revisions to these documents will be provided
- 972 to the IRB by the investigator, as allowable by local regulations. The principal investigator will
- ensure that the study will be conducted according to the protocol and all applicable regulations.
- 974 The protection of each subject's rights and welfare will be maintained.

#### 975 **9.13 Retention of records**

- 976 FDA regulations (21 CFR § 312.62[c]) and the ICH Guideline for GCP (see Section 4.9 of the
- 977 quideline) require that records and documents pertaining to the conduct of clinical trials and the
- 978 distribution of investigational drug, patient records, consent forms, laboratory test results, and
- 979 medication inventory records, must be retained for 2 years after the last marketing application
- 980 approval in an ICH region or after at least 2 years have elapsed since formal discontinuation of
- 981 clinical development of the investigational product. All state and local laws for retention of
- 982 records also apply.

986

987

- 983 For studies conducted outside the United States under a U.S. IND, the Principal Investigator
- 984 must comply with the record retention requirements set forth in the FDA IND regulations and the
- 985 relevant national and local health authorities, whichever is longer.

#### 10 STATISTICAL METHODS

#### 10.1 Study Design and Sample Size Justification

- 988 The primary objective of this single center, single arm phase II study is to determine the efficacy
- 989 of letermovir prophylaxis in PLL, CLL, PTCL or CTCL patients treated with alemtuzumab. The
- 990 efficacy will be measured through the CMV reactivation rate during letermovir prophylaxis (3

991 months after completion of alemtuzumab therapy). All eligible patients who receive any

992 letermovir will be included in the safety analysis, and all patients who receive ≥90% of planned

993 letermovir doses are evaluable for the efficacy analysis.

994 Fleming's two-stage design[80] will be followed to conduct the study. Previous trials reported

995 CMV reactivation rate of 30% in a similar patient population, and our own institutional data

996 revealed a similar pattern. Based on these data, we determined that a CMV reactivation rate of

- 997 30% or higher is not acceptable, which leads to our null hypothesis of a 70% safety rate. In a
- 998 pivotal phase 3 trial, letermovir prophylaxis resulted in a clinically significant 23.1% absolute
- 999 reduction (61.6% relative risk reduction) in CMV infection rate compared with placebo in
- recipients of allogeneic hematopoietic stem cell transplantation without evidence of hematologic
- toxicity [67]. Therefore, we hypothesized that letermovir prophylaxis will reduce the CMV by
- 1002 20% in our patient population to a 10% reactivation rate, which translates to an alternative
- 1003 hypothesis of 90% safety rate.
- 1004 With a one-sided type I error rate of 5% and 85% power, Fleming's two-stage design allows a
- first-stage analysis after the first 14 patients are enrolled and evaluated. If 4 or more patients
- 1006 have CMV reactivation during letermovir prophylaxis period, the regimen will be considered
- inefficacious, and the study will be terminated early due to futility. On the other hand, if none of
- the 14 patients experiences CMV reactivation, letermovir will be declared effective in preventing
- 1009 CMV reactivation, and the study will be ended early with rejection of the null hypothesis as the
- final conclusion. If CMV infection is observed in between 1 to 3 patients among the first 14, then
- the study will continue to accrue to a total of 28 patients. By the end of the study, if at least 24
- out of the 28 patients are CMV free, we will conclude the regimen effective to warrant further
- 1013 investigation.

1019

1020

1021

1022

1023

1024

10251026

1027

1028

1029

1030

1031

1032

- To account for the possibility that some patients might not be evaluable, we will allow a 5%
- over-accrual for a total target enrollment of 30 patients. With an anticipated accrual rate of 1.5
- patients a month, the study is expected to complete enrolling for the first stage in 10 months.
- 1017 With another 7 months for the primary endpoint evaluation, the first stage will finish in about 17
- months. If the second stage were to continue, the whole study can last as long as 27 months.

#### 10.2 Analysis of Primary Objective

 For efficacy analysis, the CMV reactivation rate will be defined as the proportion of patients who experience CMV reactivation (CMV DNA by real time polymerase chain reaction >500 IU/mL) during prophylaxis period among all patients who receive ≥90% of planned letermovir doses. The rate will be provided with 95% binomial confidence interval.

#### 10.3 Analysis of Secondary Objectives

1. All eligible patients who receive any letermovir prophylaxis will be included in the tolerability analysis. Adverse event data will be described and graded per the NCI CTCAE v5.0 guidelines. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns, especially for grade 3 or above adverse events. To assess tolerability, we also capture the proportion of patients who require dose reduction as well as those who go off treatment due to adverse events.

- Clinically significant CMV reactivation be determined per the Disease Definitions
   Working Group of the Cytomegalovirus Drug Development Forum [71] (Appendix 12.1).
- 1035 3. OS of patients treated with alemtuzumab after letermovir prophylaxis will be calculated from trial enrollment to the occurrence of (death due to any cause), censoring event-free patients at time of last follow-up. OS will be estimated with the method of Kaplan-Meier (KM), where KM curves will be drawn to aid with visualization and estimates provided with 95% confidence intervals.

#### 10.4 Analysis of Exploratory Objectives

- 1041 CMV DNA Sequence Analysis to be performed only in subjects with CMV reactivation.
- 1042 Resistance to letermovir will be monitored by retrospective genotypic analysis of the CMV
- terminase gene UL56 in CMV DNA extracts from selected plasma samples collected at the time
- of diagnosed CMV reactivation. Samples will be analyzed by standard population sequencing
- technology through an established contract laboratory with validated protocols in place. If no
- mutations are noted in UL56, then genotype testing will reflex to UL51 and UL89 (less frequent
- resistance mutations have been reported in these genes).

#### 11 REFERENCES

1049

1048

1040

- 1050 1. Foss, F.M., et al., *Peripheral T-cell lymphoma*. Blood, 2011. **117**(25): p. 6756-6767.
- 1051 2. Vose, J., et al., *International peripheral T-cell and natural killer/T-cell lymphoma study:* pathology findings and clinical outcomes. J Clin Oncol, 2008. **26**(25): p. 4124-30.
- Morgensztern, D., et al., *Lack of survival improvement in patients with peripheral T-cell lymphoma: a Surveillance, Epidemiology, and End Results analysis.* Leuk Lymphoma, 2011. **52**(2): p. 194-204.
- Weisenburger, D.D., et al., *Peripheral T-cell lymphoma, not otherwise specified: a report* of 340 cases from the International Peripheral T-cell Lymphoma Project. Blood, 2011. **117**(12): p. 3402-8.
- 1059 5. Abouyabis, A.N., et al., *Incidence and outcomes of the peripheral T-cell lymphoma subtypes in the United States.* Leuk Lymphoma, 2008. **49**(11): p. 2099-107.
- 1061 6. Morton, L.M., et al., *Lymphoma incidence patterns by WHO subtype in the United* 1062 States, 1992-2001. Blood, 2006. **107**(1): p. 265-76.
- Hristov, A.C., T. Tejasvi, and R.A. Wilcox, *Mycosis fungoides and Sezary syndrome:* 2019 update on diagnosis, risk-stratification, and management. Am J Hematol, 2019. **94**(9): p. 1027-1041.
- Agar, N.S., et al., Survival outcomes and prognostic factors in mycosis fungoides/Sezary syndrome: validation of the revised International Society for Cutaneous
   Lymphomas/European Organisation for Research and Treatment of Cancer staging proposal. J Clin Oncol, 2010. 28(31): p. 4730-9.
- Duvic, M., et al., Bexarotene is effective and safe for treatment of refractory advancedstage cutaneous T-cell lymphoma: multinational phase II-III trial results. J Clin Oncol, 2001. **19**(9): p. 2456-71.
- 10. Olsen, E.A., et al., *Phase IIb multicenter trial of vorinostat in patients with persistent,* progressive, or treatment refractory cutaneous *T-cell lymphoma*. J Clin Oncol, 2007. **25**(21): p. 3109-15.
- 1076 11. Mann, B.S., et al., *Vorinostat for treatment of cutaneous manifestations of advanced primary cutaneous T-cell lymphoma*. Clin Cancer Res, 2007. **13**(8): p. 2318-22.

- 1078 12. Whittaker, S.J., et al., *Final results from a multicenter, international, pivotal study of romidepsin in refractory cutaneous T-cell lymphoma.* J Clin Oncol, 2010. **28**(29): p. 4485-91.
- 1081 13. Piekarz, R.L., et al., *Phase II Multi-Institutional Trial of the Histone Deacetylase Inhibitor* 1082 *Romidepsin As Monotherapy for Patients With Cutaneous T-Cell Lymphoma*. Journal of 1083 Clinical Oncology, 2009. **27**(32): p. 5410-5417.
- 1084 14. Prince, H.M., et al., *Brentuximab vedotin or physician's choice in CD30-positive*1085 cutaneous T-cell lymphoma (ALCANZA): an international, open-label, randomised,
  1086 phase 3, multicentre trial. Lancet, 2017. **390**(10094): p. 555-566.
- 1087 15. Kim, Y.H., et al., *Mogamulizumab versus vorinostat in previously treated cutaneous T-cell lymphoma (MAVORIC): an international, open-label, randomised, controlled phase 3 trial.* Lancet Oncol, 2018. **19**(9): p. 1192-1204.
- 1090 16. Matutes, E., et al., *Clinical and laboratory features of 78 cases of T-prolymphocytic leukemia.* Blood, 1991. **78**(12): p. 3269-74.
- 1092 17. Sud, A. and C. Dearden, *T-cell Prolymphocytic Leukemia*. Hematol Oncol Clin North Am, 2017. **31**(2): p. 273-283.
- 1094 18. Dearden, C.E., et al., *Alemtuzumab therapy in T-cell prolymphocytic leukemia:*1095 comparing efficacy in a series treated intravenously and a study piloting the
  1096 subcutaneous route. Blood, 2011. **118**(22): p. 5799-802.
- 1097 19. Pawson, R., et al., *Treatment of T-cell prolymphocytic leukemia with human CD52 antibody.* J Clin Oncol, 1997. **15**(7): p. 2667-72.
- 1099 20. Ferrajoli, A., et al., *Phase II study of alemtuzumab in chronic lymphoproliferative disorders.* Cancer, 2003. **98**(4): p. 773-8.
- 1101 21. Keating, M.J., et al., Campath-1H treatment of T-cell prolymphocytic leukemia in patients for whom at least one prior chemotherapy regimen has failed. J Clin Oncol, 2002. **20**(1): p. 205-13.
- 1104 22. Dearden, C.E., et al., *High remission rate in T-cell prolymphocytic leukemia with* 1105 *CAMPATH-1H.* Blood, 2001. **98**(6): p. 1721-6.
- 1106 23. Krishnan, B., et al., Stem cell transplantation after alemtuzumab in T-cell prolymphocytic
   1107 leukaemia results in longer survival than after alemtuzumab alone: a multicentre
   1108 retrospective study. Br J Haematol, 2010. 149(6): p. 907-10.
- 1109 24. Wiktor-Jedrzejczak, W., et al., Hematopoietic stem cell transplantation in T 1110 prolymphocytic leukemia: a retrospective study from the European Group for Blood and
   1111 Marrow Transplantation and the Royal Marsden Consortium. Leukemia, 2012. 26(5): p.
   1112 972-6.
- 1113 25. Guillaume, T., et al., *Allogeneic hematopoietic stem cell transplantation for T-*1114 prolymphocytic leukemia: a report from the French society for stem cell transplantation
  1115 (SFGM-TC). Eur J Haematol, 2015. **94**(3): p. 265-9.
- 1116 26. Kalaycio, M.E., et al., *Allogeneic hematopoietic cell transplant for prolymphocytic leukemia*. Biol Blood Marrow Transplant, 2010. **16**(4): p. 543-7.
- 1118 27. Poggio, T., J. Duyster, and A. Illert, *Current Immunotherapeutic Approaches in T Cell Non-Hodgkin Lymphomas.* Cancers, 2018. **10**(9): p. 339.
- 1120 28. Enblad, G., et al., *A pilot study of alemtuzumab (anti-CD52 monoclonal antibody)*1121 therapy for patients with relapsed or chemotherapy-refractory peripheral *T-cell*1122 lymphomas. Blood, 2004. **103**(8): p. 2920-4.
- Stewart, J.R., et al., Alemtuzumab is an effective third-line treatment versus single-agent gemcitabine or pralatrexate for refractory Sezary syndrome: a systematic review. Eur J Dermatol, 2018. 28(6): p. 764-774.
- 1126 30. Bernengo, M.G., et al., *Low-dose intermittent alemtuzumab in the treatment of Sezary*1127 syndrome: clinical and immunologic findings in 14 patients. Haematologica, 2007. **92**(6):
  1128 p. 784-94.

- 1129 31. Watanabe, R., et al., *Alemtuzumab therapy for leukemic cutaneous T-cell lymphoma:*1130 *diffuse erythema as a positive predictor of complete remission.* JAMA Dermatol, 2014.
  1131 **150**(7): p. 776-9.
- 1132 32. Kluin-Nelemans, H.C., et al., *Intensified alemtuzumab-CHOP therapy for peripheral T-cell lymphoma*. Ann Oncol, 2011. **22**(7): p. 1595-600.
- 1134 33. Roswarski, J., et al., *Phase 1/2 study of alemtuzumab with dose-adjusted EPOCH in untreated aggressive T and NK cell lymphomas.* Leuk Lymphoma, 2019. **60**(8): p. 2062-1136 2066.
- 1137 34. Ravandi, F., et al., *Phase II study of alemtuzumab in combination with pentostatin in patients with T-cell neoplasms.* J Clin Oncol, 2009. **27**(32): p. 5425-30.
- 1139 35. Cannon, M.J., D.S. Schmid, and T.B. Hyde, *Review of cytomegalovirus seroprevalence* 1140 and demographic characteristics associated with infection. Rev Med Virol, 2010. **20**(4): 1141 p. 202-13.
- 1142 36. Borst, E.M., et al., *The human cytomegalovirus UL51 protein is essential for viral*1143 *genome cleavage-packaging and interacts with the terminase subunits pUL56 and*1144 *pUL89.* J Virol, 2013. **87**(3): p. 1720-32.
- 1145 37. Boeckh, M., et al., *Cytomegalovirus in hematopoietic stem cell transplant recipients:*1146 *Current status, known challenges, and future strategies.* Biol Blood Marrow Transplant,
  1147 2003. **9**(9): p. 543-58.
- 1148 38. El Chaer, F., D.P. Shah, and R.F. Chemaly, *How I treat resistant cytomegalovirus*1149 *infection in hematopoietic cell transplantation recipients.* Blood, 2016. **128**(23): p. 26241150 2636.
- Allice, T., et al., *Valganciclovir as pre-emptive therapy for cytomegalovirus infection post*allogenic stem cell transplantation: implications for the emergence of drug-resistant cytomegalovirus. J Antimicrob Chemother, 2009. **63**(3): p. 600-8.
- Hantz, S., et al., *Drug-resistant cytomegalovirus in transplant recipients: a French cohort study.* J Antimicrob Chemother, 2010. **65**(12): p. 2628-40.
- 1156 41. Sharma, K., et al., *Phase II Study of Alemtuzumab (CAMPATH-1) in Patients with HTLV-1-Associated Adult T-cell Leukemia/lymphoma.* Clin Cancer Res, 2017. **23**(1): p. 35-42.
- 1158 42. Kim, J.G., et al., *Alemtuzumab plus CHOP as front-line chemotherapy for patients with peripheral T-cell lymphomas: a phase II study.* Cancer Chemother Pharmacol, 2007. **60**(1): p. 129-34.
- 1161 43. Binder, C., et al., *CHO(E)P-14 followed by alemtuzumab consolidation in untreated*1162 peripheral *T cell lymphomas: final analysis of a prospective phase II trial.* Ann Hematol,
  1163 2013. **92**(11): p. 1521-8.
- Weidmann, E., et al., A phase II study of alemtuzumab, fludarabine, cyclophosphamide,
  and doxorubicin (Campath-FCD) in peripheral T-cell lymphomas. Leuk Lymphoma,
  2010. 51(3): p. 447-55.
- Hopfinger, G., et al., Sequential chemoimmunotherapy of fludarabine, mitoxantrone, and cyclophosphamide induction followed by alemtuzumab consolidation is effective in T-cell prolymphocytic leukemia. Cancer, 2013. **119**(12): p. 2258-67.
- Kuan, J.W., et al., The Outcome of HyperCVAD Combined with Alemtuzumab for the
   Treatment of Aggressive T-Cell and NK-Cell Neoplasms. Indian J Hematol Blood
   Transfus, 2011. 27(3): p. 136-45.
- 1173 47. Intragumtornchai, T., et al., *Alemtuzumab in Combination with CHOP and ESHAP as*1174 First-Line Treatment in Peripheral T-Cell Lymphoma. Blood, 2006. **108**(11): p. 47401175 4740.
- 1176 48. Kim, S.J., et al., *Dose modification of alemtuzumab in combination with dexamethasone,*1177 *cytarabine, and cisplatin in patients with relapsed or refractory peripheral T-cell*1178 *lymphoma: analysis of efficacy and toxicity.* Invest New Drugs, 2012. **30**(1): p. 368-75.

- 1179 49. Rupoli, S., et al., Alemtuzumab in Combination with Interferon-α or Gemcitabine in
   1180 Aggressive and Advanced Cutaneous T-Cell Lymphomas: Report of Preliminary Results.
   1181 Blood, 2008. 112(11): p. 5000-5000.
- de Masson, A., et al., *Long-term efficacy and safety of alemtuzumab in advanced primary cutaneous T-cell lymphomas.* Br J Dermatol, 2014. **170**(3): p. 720-4.
- Dumitriu, B., et al., *Alemtuzumab in T-cell large granular lymphocytic leukaemia: interim results from a single-arm, open-label, phase 2 study.* Lancet Haematol, 2016. **3**(1): p. e22-9.
- 1187 52. Alinari, L., et al., Subcutaneous alemtuzumab for Sezary Syndrome in the very elderly. Leuk Res, 2008. **32**(8): p. 1299-303.
- 1189 53. Nguyen, D.D., et al., *Cytomegalovirus viremia during Campath-1H therapy for relapsed* 1190 and refractory chronic lymphocytic leukemia and prolymphocytic leukemia. Clin 1191 Lymphoma, 2002. **3**(2): p. 105-10.
- 1192 54. Querfeld, C., et al., Alemtuzumab for relapsed and refractory erythrodermic cutaneous 1193 T-cell lymphoma: a single institution experience from the Robert H. Lurie Comprehensive Cancer Center. Leuk Lymphoma, 2009. **50**(12): p. 1969-76.
- Zinzani, P.L., et al., *Preliminary observations of a phase II study of reduced-dose alemtuzumab treatment in patients with pretreated T-cell lymphoma*. Haematologica, 2005. **90**(5): p. 702-3.
- 1198 56. Kennedy, G.A., et al., *Treatment of patients with advanced mycosis fungoides and Sezary syndrome with alemtuzumab.* Eur J Haematol, 2003. **71**(4): p. 250-6.
- Lundin, J., et al., *Phase 2 study of alemtuzumab (anti-CD52 monoclonal antibody) in patients with advanced mycosis fungoides/Sezary syndrome.* Blood, 2003. **101**(11): p. 4267-72.
- 1203 58. Clark, R.A., et al., *Skin effector memory T cells do not recirculate and provide immune* 1204 protection in alemtuzumab-treated CTCL patients. Sci Transl Med, 2012. **4**(117): p. 1205 117ra7.
- 1206 59. Novelli, S., et al., *Alemtuzumab treatment for Sezary syndrome: A single-center* experience. J Dermatolog Treat, 2016. **27**(2): p. 179-81.
- 1208 60. Buckstein, R., et al., *Alemtuzumab and CHOP Chemotherapy for the Treatment of*1209 *Aggressive Histology Peripheral T Cell Lymphomas: A Multi-Center Phase I Study.* Clin
  1210 Lymphoma Myeloma Leuk, 2016. **16**(1): p. 18-28 e4.
- 1211 61. Kim, S.J., et al., *Alemtuzumab and DHAP (A-DHAP) is effective for relapsed peripheral*1212 *T-cell lymphoma, unspecified: interim results of a phase II prospective study.* Ann Oncol,
  1213 2009. **20**(2): p. 390-2.
- Wulf, G.G., et al., Reduced intensity conditioning and allogeneic stem cell
   transplantation after salvage therapy integrating alemtuzumab for patients with relapsed
   peripheral T-cell non-Hodgkin's lymphoma. Bone Marrow Transplant, 2005. 36(3): p.
   271-3.
- 1218 63. Beltran-Garate, B., et al., *Alemtuzumab in Patients with Advanced Mycosis Fungoides* and Sezary Syndrome. Blood, 2007. **110**(11): p. 3425-3425.
- Oliveira, A., et al., Sezary syndrome presenting with leonine facies and treated with low-dose subcutaneous alemtuzumab. Dermatol Online J, 2011. **17**(11): p. 6.
- Fernandes, I.C., et al., Can the level of CD52 expression on Sezary cells be used to predict the response of Sezary syndrome to alemtuzumab? J Am Acad Dermatol, 2012. **67**(5): p. 1083-5.
- 1225 66. Kim, S.J., et al., *Non-bacterial infections in Asian patients treated with alemtuzumab: a*1226 retrospective study of the Asian Lymphoma Study Group. Leuk Lymphoma, 2012. **53**(8):
  1227 p. 1515-24.
- 1228 67. Marty, F.M., et al., *Letermovir Prophylaxis for Cytomegalovirus in Hematopoietic-Cell* 1229 *Transplantation.* N Engl J Med, 2017. **377**(25): p. 2433-2444.

- 1230 68. Goldner, T., et al., *The novel anticytomegalovirus compound AIC246 (Letermovir)*1231 *inhibits human cytomegalovirus replication through a specific antiviral mechanism that*1232 *involves the viral terminase.* J Virol, 2011. **85**(20): p. 10884-93.
- 1233 69. Lischka, P., et al., *In vitro and in vivo activities of the novel anticytomegalovirus* compound AIC246. Antimicrob Agents Chemother, 2010. **54**(3): p. 1290-7.
- 1235 70. Ljungman, P., et al., A Mortality Analysis of Letermovir Prophylaxis for Cytomegalovirus 1236 (CMV) in CMV-Seropositive Recipients of Allogeneic Hematopoietic-Cell 1237 Transplantation. Clin Infect Dis, 2019.
- 1238 71. Ljungman, P., et al., *Definitions of Cytomegalovirus Infection and Disease in Transplant*1239 *Patients for Use in Clinical Trials: Table 1.* Clinical Infectious Diseases, 2017. **64**(1): p.
  1240 87-91.
- 1241 72. Chou, S., *A third component of the human cytomegalovirus terminase complex is involved in letermovir resistance.* Antiviral Res, 2017. **148**: p. 1-4.
- 1243 73. Lischka, P., D. Michel, and H. Zimmermann, *Characterization of Cytomegalovirus*1244 Breakthrough Events in a Phase 2 Prophylaxis Trial of Letermovir (AIC246, MK 8228). J
  1245 Infect Dis, 2016. **213**(1): p. 23-30.
- 1246 74. Chou, S., L.E. Satterwhite, and R.J. Ercolani, *New Locus of Drug Resistance in the*1247 *Human Cytomegalovirus UL56 Gene Revealed by In Vitro Exposure to Letermovir and*1248 *Ganciclovir.* Antimicrob Agents Chemother, 2018. **62**(9).
- 1249 75. Chou, S., *Rapid In Vitro Evolution of Human Cytomegalovirus UL56 Mutations That*1250 Confer Letermovir Resistance. Antimicrob Agents Chemother, 2015. **59**(10): p. 6588-93.
- 1251 76. Goldner, T., et al., *Geno- and phenotypic characterization of human cytomegalovirus*1252 *mutants selected in vitro after letermovir (AIC246) exposure.* Antimicrob Agents
  1253 Chemother, 2014. **58**(1): p. 610-3.
- 1254 77. Chou, S., Comparison of Cytomegalovirus Terminase Gene Mutations Selected after
  1255 Exposure to Three Distinct Inhibitor Compounds. Antimicrob Agents Chemother, 2017.
  1256 **61**(11).
- 1257 78. Lischka, P., et al., *Impact of glycoprotein B genotype and naturally occurring ORF UL56* 1258 polymorphisms upon susceptibility of clinical human cytomegalovirus isolates to
   1259 letermovir. Antiviral Res, 2016. 132: p. 204-9.
- T9. Goldner, T., H. Zimmermann, and P. Lischka, *Phenotypic characterization of two naturally occurring human Cytomegalovirus sequence polymorphisms located in a distinct region of ORF UL56 known to be involved in in vitro resistance to letermovir.* Antiviral Res, 2015. **116**: p. 48-50.
- 1264 80. Fleming, T.R., *One-sample multiple testing procedure for phase II clinical trials.* 1265 Biometrics, 1982. **38**(1): p. 143-51.

#### 1267 **12 APPENDICES**

1266

1268

## 12.1 CMV Disease Definitions Working Group of the Cytomegalovirus Drug

## 1269 **Development Forum**

| CMV Disease | Diagnostic criteria | Notes |
|---|---|---|
| Pneumonia | Clinical symptoms and/or signs of pneumonia such as new infiltrates on imaging, hypoxia, tachypnea, and/or dyspnea AND | PCR may be too sensitive, so<br>detection of CMV by PCR alone is<br>insufficient for the diagnosis of<br>CMV pneumonia. |

| | CMV documented in BAL or lung tissue by virus isolation, rapid culture, histopathology, IHC, or DNA hybridization techniques | <ul> <li>Detection of fungal co-pathogens like Aspergillus spp. + "halo" sign (radiology) indicates fungal, rather than CMV pneumonia.</li> <li>Superinfection or coinfection with other pathogens may occur and should be noted when present.</li> </ul> |
|---|---|---|
| GI | Upper and/or lower gastrointestinal (GI) symptoms AND macroscopic mucosal lesions AND CMV documented in tissue by histopathology, virus isolation, rapid culture, IHC, or DNA hybridization techniques. | <ul> <li>PCR may be too sensitive, so detection of CMV by PCR alone is insufficient for the diagnosis of CMV GI disease</li> <li>Studies should give information regarding the presence or absence of GI GVHD in HSCT recipients.</li> </ul> |
| Hepatitis | Abnormal liver function tests AND CMV documented in tissue by histopathology, IHC, virus isolation, rapid culture, or DNA hybridization techniques AND Absence of other documented cause of hepatitis, including DILI | Studies should give information<br>regarding the presence or<br>absence of hepatic GVHD in<br>HSCT recipients. |
| CNS | CNS symptoms AND Detection of CMV in CNS tissue by virus isolation, rapid culture, IHC, in situ hybridization, or (preferably) quantitative PCR. | Probable disease requires CNS symptoms plus detection of CMV in CSF without visible contamination of blood plus abnormal imaging results or evidence of encephalitis on electroencephalography. |
| Retinitis | Typical ophthalmological signs judged by an ophthalmologist experienced with the diagnosis of CMV retinitis OR CMV documented in vitreous fluid by NAT (for example PCR) | |
| Nephritis | Renal dysfunction AND Detection of CMV by virus isolation, rapid culture, IHS, or in situ hybridization in a kidney biopsy specimen AND Identification of histologic features of CMV infection | The detection of CMV in urine by<br>PCR or culture is not sufficient for<br>the diagnosis of CMV nephritis as<br>asymptomatic viral shedding in<br>urine is common. |

| Cystitis | Signs/symptoms of cystitis AND Detection of CMV by virus isolation, rapid culture, IHC, or in situ hybridization in a bladder biopsy specimen AND Histologic features of CMV infection. | The detection of CMV in urine by<br>PCR or culture is not sufficient for<br>the diagnosis of CMV cystitis as<br>asymptomatic viral shedding in<br>urine is common. |
|---|---|---|
| Myocarditis | Signs/symptoms of myocarditis AND Detection of CMV by virus isolation, rapid culture, IHC, or in situ hybridization in a myocardial biopsy specimen AND Histologic features of CMV infection. | |
| Pancreatitis | Signs/symptoms of myocarditis AND Detection of CMV by virus isolation, rapid culture, IHC, or in situ hybridization in a pancreatic biopsy specimen AND Histologic features of CMV infection. | |
| Other | Presence of compatible symptoms in other organs AND Detection of CMV by virus isolation, rapid culture, IHC, or in situ hybridization in a biopsy specimen | |

Reference [71]. BAL= bronchoalveolar lavage; CMV = cytomegalovirus; CNS = central nervous system; DILI = drug induced liver injury; GI = gastrointestinal; GVHD = graft versus host disease; HSCT = hematopoietic stem cell transplant; IHC = immunohistochemistry; NAT = nucleic acid testing; PCR = polymerase chain reaction

## 1271 **12.2 Eastern Cooperative Oncology Group Performance Status Scale**

1270

| ECOG | Description |
|---|---|
| 0 | Asymptomatic (Fully active, able to carry on all predisease activities without restriction) |
| 1 | Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work) |
| 2 | Symptomatic, <50% in bed during the day (Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours) |
| 3 | Symptomatic, >50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours) |
| 4 | Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair) |

| 5 | Death |
|---|-------|
|---|-------|

1272

1273

## 12.3 Child-Pugh Classification of liver disease

| | Scoring by Anomaly | | |
|---|---|---|---|
| Signs or symptom | 1 point | 2 points | 3 points |
| Hepatic encephalopathy <sup>1</sup> | Absent | Grade 1 or 2 | Grade 3 or 4 |
| Ascites | Absent | Mild | Moderate |
| Bilirubin (µmol/L) | < 2 mg/dL | 2 – 3 mg/dL | > 3 mg/dL |
| Albumin (g/dL) | > 3.5 g/dL | 2.8 – 3.5 g/dL | < 2.8 g/dL |
| Prothrombin time (INR) | < 1.7 | 1.7 – 2.3 | > 2.3 |

<sup>1</sup>Hepatic encephalopathy grading: Grade 1: Altered mood/confusion

Grade 2: Inappropriate behavior, impending stupor, somnolence

Grade 3: Markedly confused, stuporous but arousable

Grade 4: Comatose/unresponsive

1274

| Child-Pugh Score interpretation | |
|---|---|
| 5-6 points | Child-Pugh Stage A (mild hepatic insufficiency) |
| | Child-Pugh Stage B (moderate hepatic insufficiency*) |
| | Child-Pugh Stage C (severe hepatic insufficiency) |
| <b>7</b> . | mia is the only abnormality noted, the subject will need to have a score of ≥7 |

to qualify for moderate hepatic insufficiency for this study